CLINICAL TRIAL: NCT03307785
Title: Phase 1b Dose-Finding Study of Niraparib, TSR-022, Bevacizumab, and Platinum-Based Doublet Chemotherapy in Combination With TSR-042 in Patients With Advanced or Metastatic Cancer
Brief Title: Study of Niraparib, TSR-022, Bevacizumab, and Platinum-Based Doublet Chemotherapy in Combination With TSR-042
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tesaro, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 213351; 3000-01-002 (Other: Tesaro)
Record Dates: First submitted 2017-09-26; First posted 2017-10-12 (Actual); Results first posted 2021-05-10 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Neoplasms; Metastatic Cancer; Advanced Cancer; Solid Tumor; Non Small Cell Lung Cancer Metastatic; Non Small Cell Lung Cancer Stage IIIB; Non Small Cell Lung Cancer
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung | interventions — niraparib; dostarlimab; CP protocol; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Part A: TSR-042 and niraparib 200 mg QD (Experimental): Patients will receive TSR-042 500 milligram (mg), intravenous (IV) infusion on Day 1 of every cycle (every 3 weeks [Q3W]) for 4 cycles (each cycle is 21 days); followed by TSR-042 1000 mg, IV infusion on Day 1 of every other cycle (every 6 weeks [Q6W]) beginning on Day 1 of Cycle 5 along with niraparib 200 mg, once daily (QD), orally on Days 1 to 21 repeated Q3W.
  Interventions: Drug: Niraparib; Drug: TSR-042
- Part A: TSR-042 and niraparib 300 mg QD (Experimental): Patients will receive TSR-042 500 mg, IV infusion on Day 1 of every cycle (Q3W) for 4 cycles (each cycle is 21 days); followed by TSR-042 1000 mg, IV infusion on Day 1 of every other cycle (Q6W) beginning on Day 1 of Cycle 5 along with niraparib 300 mg, QD, orally on Days 1 to 21 repeated Q3W.
  Interventions: Drug: Niraparib; Drug: TSR-042
- Part B: TSR-042 and carboplatin-paclitaxel (Experimental): Patients will receive TSR-042 500 mg, IV infusion on Day 1 of every cycle (Q3W) for 4 cycles (each cycle is 21 days); followed by TSR-042 1000 mg, IV infusion on Day 1 of every other cycle (Q6W) beginning on Day 1 of Cycle 5 along with carboplatin, IV infusion on Day 1 Q3W and paclitaxel 175 milligram per square meter (mg/m^2), IV infusion on Day 1 Q3W administered for 4 to 6 cycles.
  Interventions: Drug: TSR-042; Drug: Carboplatin-Paclitaxel
- Part C: TSR-042, niraparib 200 mg QD and bevacizumab (Experimental): Patients will receive TSR-042 500 mg, IV infusion on Day 1 of every cycle (Q3W) for 4 cycles (each cycle is 21 days); followed by TSR-042 1000 mg, IV infusion on Day 1 of every other cycle (Q6W) beginning on Day 1 of Cycle 5 along with niraparib 200 mg administered orally on Days 1 to 21 repeated Q3W and bevacizumab 15 mg/kilogram (kg), IV infusion on Day 1 of every 21-day cycle Q3W for up to 15 months.
  Interventions: Drug: Niraparib; Drug: TSR-042; Drug: Bevacizumab
- Part C: TSR-042, niraparib 300 mg QD and bevacizumab (Experimental): Patients will receive TSR-042 500 mg, IV infusion on Day 1 of every cycle (Q3W) for 4 cycles (each cycle is 21 days); followed by TSR-042 1000 mg, IV infusion on Day 1 of every other cycle (Q6W) beginning on Day 1 of Cycle 5 along with niraparib 300 mg administered orally on Days 1 to 21 repeated Q3W and bevacizumab 15 mg/kg, IV infusion on Day 1 of every 21-day cycle Q3W for up to 15 months.
  Interventions: Drug: Niraparib; Drug: TSR-042; Drug: Bevacizumab
- Part D: TSR-042, carboplatin-paclitaxel and bevacizumab (Experimental): Patients will receive TSR-042 500 mg, IV infusion on Day 1 of every cycle (Q3W) for 4 cycles (each cycle is 21 days); followed by TSR-042 1000 mg, IV infusion on Day 1 of every other cycle (Q6W) beginning on Day 1 of Cycle 5 along with carboplatin, IV infusion on Day 1 Q3W and paclitaxel 175 mg/m^2, IV infusion on Day 1 Q3W administered for 4 to 6 cycles; and bevacizumab 15 mg/kg, IV infusion on Day 1 of every 21-day cycle Q3W for up to 15 months.
  Interventions: Drug: TSR-042; Drug: Carboplatin-Paclitaxel; Drug: Bevacizumab
- Part E: TSR-042 and carboplatin-pemetrexed (Experimental): Patients will receive TSR-042 500 mg, IV infusion on Day 1 of every cycle (Q3W) along with carboplatin, IV infusion on Day 1 Q3W and pemetrexed 500 mg/m^2, IV infusion on Day 1 Q3W (with vitamin supplementation) administered for 6 cycles (each cycle is 21 days).
  Interventions: Drug: TSR-042; Drug: Carboplatin-Pemetrexed
- Part F: TSR-042, TSR-022, and carboplatin-pemetrexed (Experimental): Patients will receive TSR-042 500 mg, IV infusion on Day 1 of every cycle (Q3W); and TSR-022 900 mg, IV infusion on Day 1 Q3W along with carboplatin, IV infusion on Day 1 Q3W administered for 5 cycles (each cycle is 21 days); and pemetrexed 500 mg/m^2, IV infusion on Day 1 Q3W (with vitamin supplementation).
  Interventions: Drug: TSR-042; Drug: TSR-022; Drug: Carboplatin-Pemetrexed
- Part G: TSR-042 and carboplatin-nab-paclitaxel (Experimental): Patients will receive TSR-042 500 mg, IV infusion on Day 1 of every cycle (Q3W) along with carboplatin, IV infusion on Day 1 Q3W for 4 to 6 cycles (each cycle is 21 days) and nab-paclitaxel 100 mg/m^2, IV infusion on Days 1, 8 and 15 (every week [Q1W]) of every 3 week cycle for 4 to 6 cycles.
  Interventions: Drug: TSR-042; Drug: Carboplatin-Nab-Paclitaxel
- Part H: TSR-042, TSR-022, and carboplatin-nab-paclitaxel (Experimental): Patients will receive TSR-042 500 mg, IV infusion on Day 1 of every cycle (Q3W); followed by TSR-022 900 mg, IV infusion on Day 1 Q3W along with carboplatin, IV infusion on Day 1 Q3W for 4 to 6 cycles (each cycle is 21 days) and nab-paclitaxel 100 mg/m^2, IV infusion on Days 1, 8 and 15 (Q1W) of every 3 week cycle for 4 to 6 cycles.
  Interventions: Drug: TSR-042; Drug: TSR-022; Drug: Carboplatin-Nab-Paclitaxel
- Part I: TSR-042, TSR-022, and carboplatin-paclitaxel (Experimental): Patients will receive TSR-042 500 mg, IV infusion on Day 1 of every cycle (Q3W); followed by TSR-022 900 mg, IV infusion on Day 1 Q3W along with carboplatin, IV infusion on Day 1 Q3W and paclitaxel 175 mg/m^2, IV infusion on Day 1 Q3W for 4 to 6 cycles (each cycle is 21 days).
  Interventions: Drug: TSR-042; Drug: Carboplatin-Paclitaxel; Drug: TSR-022

INTERVENTIONS:
Drug: Niraparib — Niraparib is a potent, orally active PARP1 and PARP2 inhibitor being developed as a treatment for patients with tumors that harbor defects in the homologous recombination DNA repair pathway or that are driven by PARP-mediated transcription factors.
  Other Names: Zejula
  Arms: Part A: TSR-042 and niraparib 200 mg QD; Part A: TSR-042 and niraparib 300 mg QD; Part C: TSR-042, niraparib 200 mg QD and bevacizumab; Part C: TSR-042, niraparib 300 mg QD and bevacizumab
Drug: TSR-042 — TSR-042 is a humanized monoclonal antibody that binds with high affinity to PD-1 resulting in inhibition of binding to programmed death receptor ligands 1 and 2 (PD-L1 and PD-L2).
Drug: Carboplatin-Paclitaxel — Carboplatin in combination with paclitaxel is a chemotherapy treatment that has been shown to be efficacious against a variety of different tumor types, including non-small cell lung cancer [NSCLC], ovarian cancer, endometrial cancer, and head and neck cancer.
  Arms: Part B: TSR-042 and carboplatin-paclitaxel; Part D: TSR-042, carboplatin-paclitaxel and bevacizumab; Part I: TSR-042, TSR-022, and carboplatin-paclitaxel
Drug: Bevacizumab — Bevacizumab is a chemotherapy treatment that has been shown to be efficacious against a variety of different cancer types, including colon cancer, lung cancer, glioblastoma, and renal-cell carcinoma. Bevacizumab is in the angiogenesis inhibitor and monoclonal antibody families of medication. It works by slowing the growth of new blood vessels.
  Other Names: Avastin
  Arms: Part C: TSR-042, niraparib 200 mg QD and bevacizumab; Part C: TSR-042, niraparib 300 mg QD and bevacizumab; Part D: TSR-042, carboplatin-paclitaxel and bevacizumab
Drug: TSR-022 — TSR-022 is a monoclonal antibody against TIM-3 (also called HAVCR2), an immune checkpoint receptor. Immune checkpoint proteins are molecules that help to regulate the immune system so it does not mistakenly attack healthy cells. However, they can also keep immune cells from recognizing and killing cancer cells.
  TIM-3 is found on the surface of certain T-cells, including tumor-infiltrating T-cells, that have left the bloodstream and migrated into the tumor environment. By binding to and blocking TIM-3, TRS-022 allows for T-cells to become activated so as to enhance T-cell-mediated attacks on tumors. These attacks reduce their growth.
  Arms: Part F: TSR-042, TSR-022, and carboplatin-pemetrexed; Part H: TSR-042, TSR-022, and carboplatin-nab-paclitaxel; Part I: TSR-042, TSR-022, and carboplatin-paclitaxel
Drug: Carboplatin-Pemetrexed — Pemetrexed and platinum therapy in combination with pembrolizumab (anti-PD-1 antibody) has proven to be efficacious in a first line setting for nonsquamous NSCLC patients
  Arms: Part E: TSR-042 and carboplatin-pemetrexed; Part F: TSR-042, TSR-022, and carboplatin-pemetrexed
Drug: Carboplatin-Nab-Paclitaxel — Nab-paclitaxel is a formulation of paclitaxel that is indicated for locally advanced or metastatic NSCLC, as first-line treatment in combination with carboplatin in patients who are not candidates for curative surgery or radiation therapy. Nab-paclitaxel has shown increased ORR and time to progression in metastatic breast cancer compared with solvent-based paclitaxel and has shown antitumor activity and improved ORR compared with solvent-based paclitaxel as first-line therapy in patients with NSCLC.
  Arms: Part G: TSR-042 and carboplatin-nab-paclitaxel; Part H: TSR-042, TSR-022, and carboplatin-nab-paclitaxel

SUMMARY:
Part A: To test the safety and tolerability of combination therapy with Niraparib and TSR-042 and to establish a safe dose that will be used in a Phase 2 study.

Part B: To test the safety and tolerability of combination therapy with Carboplatin-Paclitaxel and TSR-042 and to establish a safe dose that will be used in a Phase 2 study.

Part C: To test the safety and tolerability of combination therapy with Niraparib, TSR-042 and Bevacizumab and to establish a safe dose that will be used in a Phase 2 study.

Part D: To test the safety and tolerability of combination therapy with Carboplatin-Paclitaxel, TSR-042 and Bevacizumab and to establish a safe dose that will be used in a Phase 2 study.

Part E: To test the safety and tolerability of combination therapy with Carboplatin-Pemetrexed and TSR-042 and to establish a safe dose that will be used in a Phase 2 study.

Part F: To test the safety and tolerability of combination therapy with Carboplatin-Pemetrexed, TSR-022 and TSR-042 and to establish a safe dose that will be used in a Phase 2 study.

Part G: To test the safety and tolerability of combination therapy with Carboplatin-nab-Paclitaxel, TSR-042 and to establish a safe dose that will be used in a Phase 2 study.

Part H: To test the safety and tolerability of combination therapy with Carboplatin-nab-Paclitaxel, TSR-022 and TSR-042 and to establish a safe dose that will be used in a Phase 2 study.

Part I: To test the safety and tolerability of combination therapy with Carboplatin-Paclitaxel, TSR-022 and TSR-042 and to establish a safe dose that will be used in a Phase 2 study.

ELIGIBILITY:
Inclusion Criteria:

* Patient has histologically or cytologically proven advanced (unresectable) or metastatic cancer as outlined below according to study part and disease type:
* Part A: Patients with previously treated advanced or metastatic cancer. Patient may have received no more than 4 lines of treatment for advanced or metastatic cancer. Hormonal treatment will not be considered a prior line of treatment.
* Part B: Patients with advanced or metastatic cancer for which treatment with carboplatin-paclitaxel is considered appropriate therapy. Patient may have received no more than 1 prior line of chemotherapy in the metastatic setting. Hormonal treatment will not be considered a prior line of treatment.
* Part C: Patients with previously treated advanced or metastatic cancer. Patient may have received no more than 4 lines of treatment for advanced or metastatic cancer. Hormonal treatment will not be considered a prior line of treatment.
* Part D: Patients in whom carboplatin-paclitaxel and bevacizumab is considered appropriate therapy. Patient may have received no more than 1 prior line of chemotherapy in the metastatic setting. Hormonal treatment will not be considered a prior line of treatment.
* Part E and F: Patients who have not received prior systemic therapy, including targeted therapy and biologic agents, for their advanced or metastatic (Stage ≥ IIIB or IV) Non-Squamous NSCLC. Patients who have received neoadjuvant or adjuvant therapy are eligible as long as development of advanced or metastatic disease occurred at least 12 months after completion of neoadjuvant or adjuvant therapy.
* Part G, H, and I: Patients who have not received prior systemic therapy, including targeted therapy and biologic agents, for their advanced or metastatic (Stage ≥ IIIB or IV) NSCLC. Patients who have received neoadjuvant or adjuvant therapy are eligible as long as development of advanced or metastatic disease occurred at least 12 months after completion of neoadjuvant or adjuvant therapy.
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Patient has adequate organ function.
* Female patient has a negative serum pregnancy test within 72 hours prior to taking study treatment if of childbearing potential and agrees to abstain from activities that could result in pregnancy from screening through 180 days after the last dose of study treatment, or is of non-childbearing potential.
* Male patient agrees to use an adequate method of contraception and not donate sperm starting with the first dose of study treatment through 90 days after the last dose of study treatment. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient.
* Patient has measurable lesions by RECIST v1.1.

For Part A and C, in addition to the general inclusion criteria, patients must also meet the following additional criterion to be considered eligible to participate in this study:

* Patient is able to take oral medications.
* For patients to be eligible for any parts of the study using niraparib 300 mg as a starting dose, a screening actual body weight ≥ 77 kg and screening platelet count ≥ 150,000 u/L is necessary.

Exclusion Criteria: (Patients will not be eligible for the study entry if any of the following criteria are met)

* Patient has known active central nervous system metastases, carcinomatous meningitis, or both.
* Patient has a known additional malignancy that progressed or required active treatment within the last 2 years. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer.
* Patient is considered a poor medical risk due to a serious, uncontrolled medical disorder, nonmalignant systemic disease, or active infection that requires systemic therapy.
* Patient has a condition (such as transfusion-dependent anemia or thrombocytopenia), therapy, or laboratory abnormality that might confound the study results or interfere with the patient's participation
* Patient is pregnant or expecting to conceive children within the projected duration of the study, starting with the screening visit through 180 days after the last dose of study treatment.

Note: No data are available regarding the presence of niraparib or its metabolites in human milk, or on its effects on the breastfed infant or milk production. Because of the potential for serious adverse reactions in breastfed infants from niraparib, female patients should not breastfeed during treatment with niraparib and for 1 month after receiving the final dose.

* Patient has a known history of human immunodeficiency virus (type 1 or 2 antibodies).
* Patient has known active hepatitis B or hepatitis C.
* Patient has an active autoimmune disease that has required systemic treatment in the past 2 years.
* Patient has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 including ipilimumab), or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
* Patient has undergone prior treatment with a known PARP inhibitor.
* Known history or current diagnosis of MDS or AML.
* Patient has a known hypersensitivity to TSR-042 components or excipients.

For Parts B, D, E, F, G, H, and I, patients will not be eligible for study entry if any of the following additional exclusion criterion are met:

• Patient has a known hypersensitivity to any of the following relevant study treatments: carboplatin, paclitaxel, pemetrexed, nab-paclitaxel, or TSR-022 components or excipients.

For Parts C and D only, patients will not be eligible for study entry if the following additional exclusion criterion is met:

* Patient has clinically significant cardiovascular disease (e.g., significant cardiac conduction abnormalities, uncontrolled hypertension, myocardial infarction, cardiac arrhythmia or unstable angina, New York Heart Association Grade 2 or greater congestive heart failure, serious cardiac arrhythmia requiring medication, Grade 2 or greater peripheral vascular disease, and history of cerebrovascular accident [CVA]) within 6 months of enrollment.
* Patient has a history of bowel obstruction, including subocclusive disease, related to the underlying disease and history of abdominal fistula, gastrointestinal perforation, or intra abdominal abscesses. Evidence of recto-sigmoid involvement by pelvic examination or bowel involvement on CT scan or clinical symptoms of bowel obstruction.
* Patient has proteinuria as demonstrated by urine protein: creatinine ratio ≥1.0 at screening or urine dipstick for proteinuria ≥2 (patients discovered to have ≥2 proteinuria on dipstick at baseline should undergo 24-hour urine collection and must demonstrate <2 g of protein in 24 hours to be eligible).
* Patient is at increased bleeding risk due to concurrent conditions (e.g., major injuries or surgery within the past 28 days prior to start of study treatment, history of hemorrhagic stroke, transient ischemic attack, subarachnoid hemorrhage, or clinically significant hemorrhage within the past 3 months).
* Patient has a known hypersensitivity to bevacizumab components or excipients.

For Parts E and F only, patients will not be eligible for study entry if any of the following additional exclusion criteria are met:

* Patient is unable to interrupt aspirin or other nonsteroidal ant-inflammatory drugs, other than an aspirin dose ≤ 1.3 g per day, for a 5-day period (8-day period for long -acting agents, such as piroxicam.
* Patient is unable or unwilling to take folic acid, vitamin B12 supplement.
* Patient has symptomatic ascites or pleural effusion. A patient who is clinically stable following treatment for these conditions (including therapeutic thoraco- or paracentesis) is eligible.

For Parts G, H, and I only, patients will not be eligible for study entry if any of the following additional exclusion criteria are met:

• Patient has pre-existing peripheral neuropathy that is Grade ≥ 2 by Common Terminology Criteria for Adverse Events (CTCAE) version 4 criteria.

For Parts E, F, G, H and I only, patients will not be eligible for study entry if any of the following additional exclusion criteria are met:

• Patient has interstitial lung disease or a history of pneumonitis that required oral or intravenous glucocorticoids to assist with management.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2024-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- United States (8):
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Encinitas, California
  - GSK Investigational Site, San Marcos, California
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yap TA, Bessudo A, Hamilton E, Sachdev J, Patel MR, Rodon J, Evilevitch L, Duncan M, Guo W, Kumar S, Lu S, Dezube BJ, Gabrail N. IOLite: phase 1b trial of doublet/triplet combinations of dostarlimab with niraparib, carboplatin-paclitaxel, with or without bevacizumab in patients with advanced cancer. J Immunother Cancer. 2022 Mar;10(3):e003924. doi: 10.1136/jitc-2021-003924. PMID 35332062

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 60 participants were enrolled in the study and 2 participants who originally signed inform consent form (ICF) withdrew their consent shortly from study before treatment assignment and a total of 58 participants were part of the study.
Pre-assignment Details: The study consisted of two phases - Main Study Phase and Post Analysis Continued Treatment (PACT) Phase. Main Study Phase was planned to be a nine-part study with Parts A to I. However, Parts G, H and I were not initiated due to business strategic reason. In PACT phase those participants benefiting from treatment continued to receive study drug until discontinuation or withdrawal from study.
Groups:
- Main Study: Part A: TSR-042 and Niraparib 200 mg QD: Participants received TSR-042 500 milligram (mg), intravenous (IV) infusion on Day 1 of every cycle (every 3 weeks [Q3W]) for 4 cycles (each cycle was of 21 days); followed by TSR-042 1000 mg, IV infusion on Day 1 of every other cycle (every 6 weeks [Q6W]) beginning on Day 1 of Cycle 5 along with niraparib 200 mg, once daily (QD), orally on Days 1 to 21 repeated Q3W.
- Main Study: Part A: TSR-042 and Niraparib 300 mg QD: Participants received TSR-042 500 mg, IV infusion on Day 1 of every cycle (Q3W) for 4 cycles (each cycle was of 21 days); followed by TSR-042 1000 mg, IV infusion on Day 1 of every other cycle (Q6W) beginning on Day 1 of Cycle 5 along with niraparib 300 mg, QD, orally on Days 1 to 21 repeated Q3W.
- Main Study: Part B: TSR-042 and Carboplatin-paclitaxel; PACT Phase: Part B: TSR-042 and Carboplatin-paclitaxel: Participants received TSR-042 500 mg, IV infusion on Day 1 of every cycle (Q3W) for 4 cycles (each cycle was of 21 days); followed by TSR-042 1000 mg, IV infusion on Day 1 of every other cycle (Q6W) beginning on Day 1 of Cycle 5 along with carboplatin, IV infusion on Day 1 Q3W and paclitaxel 175 milligram per square meter (mg/m^2), IV infusion on Day 1 Q3W administered for 4 to 6 cycles.
- Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab: Participants received TSR-042 500 mg, IV infusion on Day 1 of every cycle (Q3W) for 4 cycles (each cycle was of 21 days); followed by TSR-042 1000 mg, IV infusion on Day 1 of every other cycle (Q6W) beginning on Day 1 of Cycle 5 along with niraparib 200 mg administered orally on Days 1 to 21 repeated Q3W and bevacizumab 15 mg/kilogram (kg), IV infusion on Day 1 of every 21-day cycle Q3W for up to 15 months.
- Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab: Participants received TSR-042 500 mg, IV infusion on Day 1 of every cycle (Q3W) for 4 cycles (each cycle was of 21 days); followed by TSR-042 1000 mg, IV infusion on Day 1 of every other cycle (Q6W) beginning on Day 1 of Cycle 5 along with niraparib 300 mg administered orally on Days 1 to 21 repeated Q3W and bevacizumab 15 mg/kg, IV infusion on Day 1 of every 21-day cycle Q3W for up to 15 months.
- Main Study: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab; PACT Phase: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab: Participants received TSR-042 500 mg, IV infusion on Day 1 of every cycle (Q3W) for 4 cycles (each cycle was of 21 days); followed by TSR-042 1000 mg, IV infusion on Day 1 of every other cycle (Q6W) beginning on Day 1 of Cycle 5 along with carboplatin, IV infusion on Day 1 Q3W and paclitaxel 175 mg/m^2, IV infusion on Day 1 Q3W administered for 4 to 6 cycles; and bevacizumab 15 mg/kg, IV infusion on Day 1 of every 21-day cycle Q3W for up to 15 months.
- Main Study: Part E: TSR-042 and Carboplatin-pemetrexed: Participants received TSR-042 500 mg, IV infusion on Day 1 of every cycle (Q3W) along with carboplatin, IV infusion on Day 1 Q3W and pemetrexed 500 mg/m^2, IV infusion on Day 1 Q3W (with vitamin supplementation) administered for approximately 6 cycles (each cycle was of 21 days).
- Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed: Participants received TSR-042 500 mg, IV infusion on Day 1 of every cycle (Q3W); and TSR-022 900 mg, IV infusion on Day 1 Q3W along with carboplatin, IV infusion on Day 1 Q3W administered for approximately 5 cycles (each cycle was of 21 days); and pemetrexed 500 mg/m^2, IV infusion on Day 1 Q3W (with vitamin supplementation).
- Main Study: Part G: TSR-042 and Carboplatin-nab-paclitaxel: Participants were planned to receive TSR-042 500 mg, IV infusion on Day 1 of every cycle (Q3W) along with carboplatin, IV infusion on Day 1 Q3W for 4 to 6 cycles (each cycle was of 21 days) and nab-paclitaxel 100 mg/m^2, IV infusion on Days 1, 8 and 15 (every week [Q1W]) of every 3 week cycle for 4 to 6 cycles.
- Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel: Participants were planned to receive TSR-042 500 mg, IV infusion on Day 1 of every cycle (Q3W); followed by TSR-022 900 mg, IV infusion on Day 1 Q3W along with carboplatin, IV infusion on Day 1 Q3W for 4 to 6 cycles (each cycle was of 21 days) and nab-paclitaxel 100 mg/m^2, IV infusion on Days 1, 8 and 15 (Q1W) of every 3 week cycle for 4 to 6 cycles.
- Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel: Participants were planned to receive TSR-042 500 mg, IV infusion on Day 1 of every cycle (Q3W); followed by TSR-022 900 mg, IV infusion on Day 1 Q3W along with carboplatin, IV infusion on Day 1 Q3W and paclitaxel 175 mg/m^2, IV infusion on Day 1 Q3W for 4 to 6 cycles (each cycle was of 21 days).
Period: Main Study: Part A: Up to 28.5 Months
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD | Main Study: Part B: TSR-042 and Carboplatin-paclitaxel | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab | Main Study: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab | Main Study: Part E: TSR-042 and Carboplatin-pemetrexed | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed | Main Study: Part G: TSR-042 and Carboplatin-nab-paclitaxel | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel | PACT Phase: Part B: TSR-042 and Carboplatin-paclitaxel | PACT Phase: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab
Started | 16 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 16 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Disease progression | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: MainStudy: PartB: Up to Approx.66months
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD | Main Study: Part B: TSR-042 and Carboplatin-paclitaxel | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab | Main Study: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab | Main Study: Part E: TSR-042 and Carboplatin-pemetrexed | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed | Main Study: Part G: TSR-042 and Carboplatin-nab-paclitaxel | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel | PACT Phase: Part B: TSR-042 and Carboplatin-paclitaxel | PACT Phase: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab
Started | 0 | 0 | 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Disease progression | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Transitioned to PACT phase | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: MainStudy: PartC:Up to Approx.60months
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD | Main Study: Part B: TSR-042 and Carboplatin-paclitaxel | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab | Main Study: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab | Main Study: Part E: TSR-042 and Carboplatin-pemetrexed | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed | Main Study: Part G: TSR-042 and Carboplatin-nab-paclitaxel | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel | PACT Phase: Part B: TSR-042 and Carboplatin-paclitaxel | PACT Phase: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab
Started | 0 | 0 | 0 | 6 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 6 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 2 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Went on Another Clinical Trial | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: MainStudy:PartD:Up to Approx. 62.5months
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD | Main Study: Part B: TSR-042 and Carboplatin-paclitaxel | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab | Main Study: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab | Main Study: Part E: TSR-042 and Carboplatin-pemetrexed | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed | Main Study: Part G: TSR-042 and Carboplatin-nab-paclitaxel | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel | PACT Phase: Part B: TSR-042 and Carboplatin-paclitaxel | PACT Phase: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab
Started | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Transitioned to PACT phase | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Completed EOT and Began New Study | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Main Study: Part E: Up to 4.4 Months
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD | Main Study: Part B: TSR-042 and Carboplatin-paclitaxel | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab | Main Study: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab | Main Study: Part E: TSR-042 and Carboplatin-pemetrexed | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed | Main Study: Part G: TSR-042 and Carboplatin-nab-paclitaxel | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel | PACT Phase: Part B: TSR-042 and Carboplatin-paclitaxel | PACT Phase: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab
Started | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Main Study: Part F: Up to 3.5 Months
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD | Main Study: Part B: TSR-042 and Carboplatin-paclitaxel | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab | Main Study: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab | Main Study: Part E: TSR-042 and Carboplatin-pemetrexed | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed | Main Study: Part G: TSR-042 and Carboplatin-nab-paclitaxel | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel | PACT Phase: Part B: TSR-042 and Carboplatin-paclitaxel | PACT Phase: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Main Study: Part G: Up to 24 Months
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD | Main Study: Part B: TSR-042 and Carboplatin-paclitaxel | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab | Main Study: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab | Main Study: Part E: TSR-042 and Carboplatin-pemetrexed | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed | Main Study: Part G: TSR-042 and Carboplatin-nab-paclitaxel | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel | PACT Phase: Part B: TSR-042 and Carboplatin-paclitaxel | PACT Phase: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Main Study: Part H: Up to 24 Months
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD | Main Study: Part B: TSR-042 and Carboplatin-paclitaxel | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab | Main Study: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab | Main Study: Part E: TSR-042 and Carboplatin-pemetrexed | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed | Main Study: Part G: TSR-042 and Carboplatin-nab-paclitaxel | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel | PACT Phase: Part B: TSR-042 and Carboplatin-paclitaxel | PACT Phase: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Main Study: Part I: Up to 24 Months
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD | Main Study: Part B: TSR-042 and Carboplatin-paclitaxel | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab | Main Study: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab | Main Study: Part E: TSR-042 and Carboplatin-pemetrexed | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed | Main Study: Part G: TSR-042 and Carboplatin-nab-paclitaxel | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel | PACT Phase: Part B: TSR-042 and Carboplatin-paclitaxel | PACT Phase: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: PACT Phase: Up to 19 Months
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD | Main Study: Part B: TSR-042 and Carboplatin-paclitaxel | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab | Main Study: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab | Main Study: Part E: TSR-042 and Carboplatin-pemetrexed | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed | Main Study: Part G: TSR-042 and Carboplatin-nab-paclitaxel | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel | PACT Phase: Part B: TSR-042 and Carboplatin-paclitaxel | PACT Phase: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (Participants transitioned from main study phase to PACT Phase.) | 1 (Participants transitioned from main study phase to PACT Phase.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Parts G, H and I were not initiated due to business strategic reason. Hence, no participants were enrolled in Parts G, H and I.
Groups:
- Total: Total of all reporting groups
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD | Main Study: Part B: TSR-042 and Carboplatin-paclitaxel | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab | Main Study: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab | Main Study: Part E: TSR-042 and Carboplatin-pemetrexed | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed | Main Study: Part G: TSR-042 and Carboplatin-nab-paclitaxel | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel | Total
Number analyzed (Participants) | 16 | 6 | 14 | 6 | 7 | 6 | 2 | 1 | 0 | 0 | 0 | 58
Age, Customized [Count of Participants; unit: Participants]
  18-64 years | 8 | 3 | 5 | 4 | 6 | 2 | 1 | 1 | 0 | 0 | 0 | 30
  65-74 years | 6 | 1 | 4 | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 17
  >=75 years | 2 | 2 | 5 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 2 | 8 | 4 | 7 | 5 | 0 | NA — Data is not reported due to participant confidentiality and privacy concerns. | 0 | 0 | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | 7 | 4 | 6 | 2 | 0 | 1 | 2 | NA — Data is not reported due to participant confidentiality and privacy concerns. | 0 | 0 | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 1 | 1 | 0 | 2 | 0 | 1 | NA — Data is not reported due to participant confidentiality and privacy concerns. | 0 | 0 | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.
  White | 16 | 5 | 13 | 6 | 5 | 6 | 1 | NA — Data is not reported due to participant confidentiality and privacy concerns. | 0 | 0 | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Dose-limiting Toxicity (DLT)
Description: An event was considered a DLT if it occurred within the first 21 days of treatment, and met one of following DLT criteria:hematologic toxicity- Grade4 thrombocytopenia persists for >=7 days from the time of adverse event(AE) onset, Grade 4 neutropenia, Grade 4 or Grade 3 febrile neutropenia persists for >=7 days, Grade4 or Grade3 anemia requiring blood transfusion, Grade 3 thrombocytopenia associated with clinically significant bleeding, Grade 3 neutropenia associated with infection as described in Common Terminology Criteria for Adverse Events (CTCAE) version 4.0, drug related Grade 3 or 4 non-hematologic toxicity, drug related Grade 3 or 4 nonhematologic laboratory abnormality if any of the following also occur: abnormality leads to hospitalization and abnormality persists for >=7 days from the time of AE onset; drug related toxicity leading to prolonged delay (>2 weeks) in initiating Cycle 2. DLTs were collected during first cycle to establish recommended phase 2 dose (RP2D).
Time Frame: 21 days
Population: Safety Population consisted of all participants who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD
Number analyzed (Participants) | 16 | 6
Participants | 2 | 0

2. Primary Outcome: Part B: Number of Participants With DLT
Description: An event was considered a DLT if it occurred within the first 21 days of treatment, and met one of following DLT criteria:hematologic toxicity- Grade4 thrombocytopenia persists for >=7 days from the time of AE onset, Grade 4 neutropenia, Grade 4 or Grade 3 febrile neutropenia persists for >=7 days, Grade4 or Grade3 anemia requiring blood transfusion, Grade 3 thrombocytopenia associated with clinically significant bleeding, Grade 3 neutropenia associated with infection as described in CTCAE version 4.0, drug related Grade 3 or 4 non-hematologic toxicity, drug related Grade 3 or 4 nonhematologic laboratory abnormality if any of the following also occur: abnormality leads to hospitalization and abnormality persists for >=7 days from the time of AE onset; drug related toxicity leading to prolonged delay (>2 weeks) in initiating Cycle 2. DLTs were collected during first cycle to establish RP2D.
Time Frame: 21 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Part B: TSR-042 and Carboplatin-paclitaxel
Number analyzed (Participants) | 14
Participants | 1

3. Primary Outcome: Part C: Number of Participants With DLT
Description: as for outcome 2
Time Frame: 21 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab
Number analyzed (Participants) | 6 | 7
Participants | 1 | 1

4. Primary Outcome: Part D: Number of Participants With DLT
Description: as for outcome 2
Time Frame: 21 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab
Number analyzed (Participants) | 6
Participants | 0

5. Primary Outcome: Part E: Number of Participants With DLT
Description: as for outcome 2
Time Frame: 21 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Part E: TSR-042 and Carboplatin-pemetrexed
Number analyzed (Participants) | 2
Participants | 0

6. Primary Outcome: Part F: Number of Participants With DLT
Description: as for outcome 2
Time Frame: 21 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed
Number analyzed (Participants) | 1
Participants | 0

7. Primary Outcome: Part G: Number of Participants With DLT
Description: An event was considered a DLT if it occurred within the first 21 days of treatment, and met one of following DLT criteria:hematologic toxicity- Grade4 thrombocytopenia persists for >=7 days from the time of AE onset, Grade 4 neutropenia, Grade 4 or Grade 3 febrile neutropenia persists for >=7 days, Grade4 or Grade3 anemia requiring blood transfusion, Grade 3 thrombocytopenia associated with clinically significant bleeding, Grade 3 neutropenia associated with infection as described in CTCAE version 4.0, drug related Grade 3 or 4 non-hematologic toxicity, drug related Grade 3 or 4 nonhematologic laboratory abnormality if any of the following also occur: abnormality leads to hospitalization and abnormality persists for >=7 days from the time of AE onset; drug related toxicity leading to prolonged delay (>2 weeks) in initiating Cycle 2. DLTs were planned to be collected during first cycle to establish RP2D.
Time Frame: 21 days
Population: Safety Population. Data was not collected as no participants were enrolled in Part G.
Arm/Group | Main Study: Part G: TSR-042 and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

8. Primary Outcome: Part H: Number of Participants With DLT
Description: as for outcome 7
Time Frame: 21 days
Population: Safety Population. Data was not collected as no participants were enrolled in Part H.
Arm/Group | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

9. Primary Outcome: Part I: Number of Participants With DLT
Description: as for outcome 7
Time Frame: 21 days
Population: Safety Population. Data was not collected as no participants were enrolled in Part I.
Arm/Group | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel
Number analyzed (Participants) | 0

10. Primary Outcome: Part A: Number of Participants With Non-serious Treatment-emergent Adverse Events (TEAEs), Serious TEAEs (STEAEs) and Adverse Events of Special Interest (AESIs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. An SAE is defined as any untoward medical occurrence that, at any dose; results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or any other situation according to medical or scientific judgement. TEAE is any event that was not present prior to the initiation of study treatment or any event already present that worsens in either intensity or frequency following exposure to study treatment. Number of participants with TEAEs, SAEs and AESIs are reported.
Time Frame: Up to 28.5 months
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD
Number analyzed (Participants) | 16 | 6
Participants
  Non-serious TEAEs | 16 | 6
  STEAEs | 11 | 4
  AESIs | 1 | 1

11. Primary Outcome: Part B: Number of Participants With Non-serious TEAEs, STEAEs and AESIs
Description: as for outcome 10
Time Frame: Up to 28.5 months
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Part B: TSR-042 and Carboplatin-paclitaxel
Number analyzed (Participants) | 14
Participants
  Non-Serious TEAEs | 14
  STEAEs | 9
  AESIs | 0

12. Primary Outcome: Part C: Number of Participants With Non-serious TEAEs, STEAEs and AESIs
Description: as for outcome 10
Time Frame: Up to 22.5 months
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab
Number analyzed (Participants) | 6 | 7
Participants
  Non-serious TEAEs | 5 | 7
  STEAEs | 3 | 3
  AESIs | 0 | 0

13. Primary Outcome: Part D: Number of Participants With Non-serious TEAEs, STEAEs and AESIs
Description: as for outcome 10
Time Frame: Up to 9.5 months
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab
Number analyzed (Participants) | 6
Participants
  Non-serious TEAEs | 6
  STEAEs | 3
  AESIs | 0

14. Primary Outcome: Part E: Number of Participants With Non-serious TEAEs, STEAEs and AESIs
Description: as for outcome 10
Time Frame: Up to 4.4 months
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Part E: TSR-042 and Carboplatin-pemetrexed
Number analyzed (Participants) | 2
Participants
  Non-serious TEAEs | 2
  STEAEs | 2
  AESIs | 0

15. Primary Outcome: Part F: Number of Participants With Non-serious TEAEs, STEAEs and AESIs
Description: as for outcome 10
Time Frame: Up to 3.5 months
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed
Number analyzed (Participants) | 1
Participants
  Non-serious TEAEs | 1
  STEAEs | 0
  AESIs | 0

16. Primary Outcome: Part G: Number of Participants With Non-serious TEAEs, STEAEs and AESIs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. An SAE is defined as any untoward medical occurrence that, at any dose; results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or any other situation according to medical or scientific judgement. TEAE is any event that was not present prior to the initiation of study treatment or any event already present that worsens in either intensity or frequency following exposure to study treatment.
Time Frame: Up to 24 months
Population: Safety Population. Data was not collected as no participants were enrolled in Part G.
Arm/Group | Main Study: Part G: TSR-042 and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

17. Primary Outcome: Part H: Number of Participants With Non-serious TEAEs, STEAEs and AESIs
Description: as for outcome 16
Time Frame: Up to 24 months
Population: Safety Population. Data was not collected as no participants were enrolled in Part H.
Arm/Group | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

18. Primary Outcome: Part I: Number of Participants With Non-serious TEAEs, STEAEs and AESIs
Description: as for outcome 16
Time Frame: Up to 24 months
Population: Safety Population. Data was not collected as no participants were enrolled in Part I.
Arm/Group | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel
Number analyzed (Participants) | 0

19. Secondary Outcome: Part A: Objective Response Rate
Description: Objective Response Rate is defined as the percentage of participants who achieved confirmed complete response (CR) or partial response (PR), evaluated using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 based on Investigator assessment; where CR=Disappearance of all target lesions. Any pathological lymph nodes must be <10 millimeters (mm) in the short axis. PR=At least a 30 percent (%) decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters.
Time Frame: Up to 28.5 months
Population: Safety Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD
Number analyzed (Participants) | 16 | 6
Percentage of participants | 25.0 | 0

20. Secondary Outcome: Part B: Objective Response Rate
Description: Objective Response Rate is defined as the percentage of participants who achieved confirmed CR or PR, evaluated using RECIST version 1.1 based on Investigator assessment; where CR=Disappearance of all target lesions. Any pathological lymph nodes must be <10 mm in the short axis. PR=At least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters.
Time Frame: Up to 28.5 months
Population: Safety Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Main Study: Part B: TSR-042 and Carboplatin-paclitaxel
Number analyzed (Participants) | 14
Percentage of participants | 42.9

21. Secondary Outcome: Part C: Objective Response Rate
Description: as for outcome 20
Time Frame: Up to 22.5 months
Population: Safety Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab
Number analyzed (Participants) | 6 | 7
Percentage of participants | 50.0 | 14.3

22. Secondary Outcome: Part D: Objective Response Rate
Description: as for outcome 20
Time Frame: Up to 9.5 months
Population: Safety Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Main Study: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab
Number analyzed (Participants) | 6
Percentage of participants | 50.0

23. Secondary Outcome: Part E: Objective Response Rate
Description: as for outcome 20
Time Frame: Up to 4.4 months
Population: Safety Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Main Study: Part E: TSR-042 and Carboplatin-pemetrexed
Number analyzed (Participants) | 2
Percentage of participants | 0

24. Secondary Outcome: Part F: Objective Response Rate
Description: as for outcome 20
Time Frame: Up to 3.5 months
Population: Safety Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed
Number analyzed (Participants) | 1
Percentage of participants | 0

25. Secondary Outcome: Part G: Objective Response Rate
Description: as for outcome 20
Time Frame: Up to 24 months
Population: Safety Population. Data was not collected as no participants were enrolled in Part G.
Arm/Group | Main Study: Part G: TSR-042 and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

26. Secondary Outcome: Part H: Objective Response Rate
Description: as for outcome 20
Time Frame: Up to 24 months
Population: Safety Population. Data was not collected as no participants were enrolled in Part H.
Arm/Group | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

27. Secondary Outcome: Part I: Objective Response Rate
Description: as for outcome 20
Time Frame: Up to 24 months
Population: Safety Population. Data was not collected as no participants were enrolled in Part I.
Arm/Group | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel
Number analyzed (Participants) | 0

28. Secondary Outcome: Part A: Duration of Response
Description: Duration of response is defined as the time from first documentation of response (CR or PR) until the time of first documentation of disease progression by RECIST version 1.1 or death by any cause.
Time Frame: Up to 28.5 months
Population: Safety Population.
Measure: Median (Full Range); unit: Months
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD
Number analyzed (Participants) | 16 | 6
Months | 7.59 [5.78 to 10.94] | NA [NA to NA] — Duration of response could not be calculated as no participants had a confirmed CR or PR in TSR-042 and niraparib 300 mg QD arm.

29. Secondary Outcome: Part B: Duration of Response
Description: as for outcome 28
Time Frame: Up to approximately 66 months
Population: Safety Population.
Measure: Median (Full Range); unit: Months
Arm/Group | Main Study: Part B: TSR-042 and Carboplatin-paclitaxel
Number analyzed (Participants) | 14
Months | NA [NA to NA] — Median and full range were not calculable due to more than 50% censored participants in this treatment group.

30. Secondary Outcome: Part C: Duration of Response
Description: as for outcome 28
Time Frame: Up to approximately 60 months
Population: Safety Population.
Measure: Median (Full Range); unit: Months
Arm/Group | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab
Number analyzed (Participants) | 6 | 7
Months | NA [NA to NA] — Median and full range were not calculable due to more than 50% censored participants in this treatment group. | NA [NA to NA] — Median and full range were not calculable due to more than 50% censored participants in this treatment group.

31. Secondary Outcome: Part D: Duration of Response
Description: as for outcome 28
Time Frame: Up to approximately 62.5 months
Population: Safety Population.
Measure: Median (Full Range); unit: Months
Arm/Group | Main Study: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab
Number analyzed (Participants) | 6
Months | NA [NA to NA] — Median and full range were not calculable due to more than 50% censored participants in this treatment group.

32. Secondary Outcome: Part E: Duration of Response
Description: as for outcome 28
Time Frame: Up to 4.4 months
Population: Safety Population.
Measure: Median (Full Range); unit: Months
Arm/Group | Main Study: Part E: TSR-042 and Carboplatin-pemetrexed
Number analyzed (Participants) | 2
Months | NA [NA to NA] — Duration of response could not be calculated as no participants had a confirmed CR or PR.

33. Secondary Outcome: Part F: Duration of Response
Description: as for outcome 28
Time Frame: Up to 3.5 months
Population: Safety Population.
Measure: Median (Full Range); unit: Months
Arm/Group | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed
Number analyzed (Participants) | 1
Months | NA [NA to NA] — Median and full range could not be calculated as there were no confirmed CR or PR.

34. Secondary Outcome: Part G: Duration of Response
Description: as for outcome 28
Time Frame: Up to 24 months
Population: Safety Population. Data was not collected as no participants were enrolled in Part G.
Arm/Group | Main Study: Part G: TSR-042 and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

35. Secondary Outcome: Part H: Duration of Response
Description: as for outcome 28
Time Frame: Up to 24 months
Population: Safety Population. Data was not collected as no participants were enrolled in Part H.
Arm/Group | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

36. Secondary Outcome: Part I: Duration of Response
Description: as for outcome 28
Time Frame: Up to 24 months
Population: Safety Population. Data was not collected as no participants were enrolled in Part I.
Arm/Group | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel
Number analyzed (Participants) | 0

37. Secondary Outcome: Part A: Disease Control Rate
Description: Disease Control Rate is defined as the percentage of participants who had achieved CR, PR, or stable disease (SD) per RECIST version 1.1.
Time Frame: Up to 28.5 months
Population: Safety Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD
Number analyzed (Participants) | 16 | 6
Percentage of participants | 43.8 | 33.3

38. Secondary Outcome: Part B: Disease Control Rate
Description: Disease Control Rate is defined as the percentage of participants who had achieved CR, PR, or SD per RECIST version 1.1.
Time Frame: Up to 28.5 months
Population: Safety Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Main Study: Part B: TSR-042 and Carboplatin-paclitaxel
Number analyzed (Participants) | 14
Percentage of participants | 57.1

39. Secondary Outcome: Part C: Disease Control Rate
Description: Disease Control Rate is defined as the percentage of participants who had achieved CR, PR, or SD per RECIST version 1.1.
Time Frame: Up to 22.5 months
Population: Safety Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab
Number analyzed (Participants) | 6 | 7
Percentage of participants | 83.3 | 85.7

40. Secondary Outcome: Part D: Disease Control Rate
Description: Disease Control Rate is defined as the percentage of participants who had achieved CR, PR, or SD per RECIST version 1.1.
Time Frame: Up to 9.5 months
Population: Safety Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Main Study: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab
Number analyzed (Participants) | 6
Percentage of participants | 83.3

41. Secondary Outcome: Part E: Disease Control Rate
Description: Disease Control Rate is defined as the percentage of participants who had achieved CR, PR, or SD per RECIST version 1.1.
Time Frame: Up to 4.4 months
Population: Safety Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Main Study: Part E: TSR-042 and Carboplatin-pemetrexed
Number analyzed (Participants) | 2
Percentage of participants | 0

42. Secondary Outcome: Part F: Disease Control Rate
Description: Disease Control Rate is defined as the percentage of participants who had achieved CR, PR, or SD per RECIST version 1.1.
Time Frame: Up to 3.5 months
Population: Safety Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed
Number analyzed (Participants) | 1
Percentage of participants | 100

43. Secondary Outcome: Part G: Disease Control Rate
Description: Disease Control Rate is defined as the percentage of participants who had achieved CR, PR, or SD per RECIST version 1.1.
Time Frame: Up to 24 months
Population: Safety Population. Data was not collected as no participants were enrolled in Part G.
Arm/Group | Main Study: Part G: TSR-042 and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

44. Secondary Outcome: Part H: Disease Control Rate
Description: Disease Control Rate is defined as the percentage of participants who had achieved CR, PR, or SD per RECIST version 1.1.
Time Frame: Up to 24 months
Population: Safety Population. Data was not collected as no participants were enrolled in Part H.
Arm/Group | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

45. Secondary Outcome: Part I: Disease Control Rate
Description: Disease Control Rate is defined as the percentage of participants who had achieved CR, PR, or SD per RECIST version 1.1.
Time Frame: Up to 24 months
Population: Safety Population. Data was not collected as no participants were enrolled in Part I.
Arm/Group | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel
Number analyzed (Participants) | 0

46. Secondary Outcome: Part A: Progression-free Survival
Description: Progression-free Survival is defined as the date of first dose to the date of disease progression or death due to any cause, whichever occurs earlier. Progressive Disease (PD) is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study.
Time Frame: Up to 28.5 months
Population: Safety Population.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD
Number analyzed (Participants) | 16 | 6
Months | 6.2 [2.2 to 9.9] | 2.8 [2.3 to 4.7]

47. Secondary Outcome: Part B: Progression-free Survival
Description: Progression-free Survival is defined as the date of first dose to the date of disease progression or death due to any cause, whichever occurs earlier. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study.
Time Frame: Up to 28.5 months
Population: Safety Population.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Main Study: Part B: TSR-042 and Carboplatin-paclitaxel
Number analyzed (Participants) | 14
Months | 17.6 [3.9 to NA] — <75% of participants experienced the event within the treatment arm. Hence, third-quartile could not be derived.

48. Secondary Outcome: Part C: Progression-free Survival
Description: as for outcome 47
Time Frame: Up to 22.5 months
Population: Safety Population.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab
Number analyzed (Participants) | 6 | 7
Months | NA [8.5 to NA] — <50% of participants experienced the event within the treatment arm. Hence, median and third-quartile could not be derived. | 9.1 [8.0 to 11.1]

49. Secondary Outcome: Part D: Progression-free Survival
Description: as for outcome 47
Time Frame: Up to 9.5 months
Population: Safety Population.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Main Study: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab
Number analyzed (Participants) | 6
Months | 7.6 [7.4 to NA] — <75% of participants experienced the event within the treatment arm. Hence, third-quartile could not be derived.

50. Secondary Outcome: Part E: Progression-free Survival
Description: as for outcome 47
Time Frame: Up to 4.4 months
Population: Safety Population.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Main Study: Part E: TSR-042 and Carboplatin-pemetrexed
Number analyzed (Participants) | 2
Months | NA [NA to NA] — Median and Inter Quartile range could not be estimated due to the low number of participants with events.

51. Secondary Outcome: Part F: Progression-free Survival
Description: as for outcome 47
Time Frame: Up to 3.5 months
Population: Safety Population.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed
Number analyzed (Participants) | 1
Months | NA [NA to NA] — Median and Inter Quartile range could not be estimated due to the low number of participant with event.

52. Secondary Outcome: Part G: Progression-free Survival
Description: Progression-free Survival is defined as the date of first dose to the date of disease progression or death due to any cause, whichever occurs earlier.
Time Frame: Up to 24 months
Population: Safety Population. Data was not collected as no participants were enrolled in Part G.
Arm/Group | Main Study: Part G: TSR-042 and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

53. Secondary Outcome: Part H: Progression-free Survival
Description: as for outcome 52
Time Frame: Up to 24 months
Population: Safety Population. Data was not collected as no participants were enrolled in Part H.
Arm/Group | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

54. Secondary Outcome: Part I: Progression-free Survival
Description: as for outcome 52
Time Frame: Up to 24 months
Population: Safety Population. Data was not collected as no participants were enrolled in Part I.
Arm/Group | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel
Number analyzed (Participants) | 0

55. Secondary Outcome: Part A: Number of Participants With Positive Anti-TSR-042 Antibodies
Description: Serum samples were collected at indicated time points and tested for the presence of antibodies that bind to TSR-042. The presence of anti-TSR-042 antibodies were assessed using a tiered approach using electrochemiluminescence (that is, screening, confirmation, titer, and neutralizing antibody assay). Anti-drug Antibody Population consisted of all participants who received at least 1 dose of study treatment and had provided a pre-dose blood sample and at least 1 post-dose blood sample at or after 96 hours.
Time Frame: Up to 28.5 months
Population: Anti-drug Antibody Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD
Number analyzed (Participants) | 16 | 6
Participants | 0 | 0

56. Secondary Outcome: Part B: Number of Participants With Positive Anti-TSR-042 Antibodies
Description: Serum samples were collected at indicated time points and tested for the presence of antibodies that bind to TSR-042. The presence of anti-TSR-042 antibodies were assessed using a tiered approach using electrochemiluminescence (that is, screening, confirmation, titer, and neutralizing antibody assay).
Time Frame: Up to 28.5 months
Population: Anti-drug Antibody Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Part B: TSR-042 and Carboplatin-paclitaxel
Number analyzed (Participants) | 14
Participants | 4

57. Secondary Outcome: Part C: Number of Participants With Positive Anti-TSR-042 Antibodies
Description: as for outcome 56
Time Frame: Up to 22.5 months
Population: Anti-drug Antibody Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab
Number analyzed (Participants) | 6 | 7
Participants | 0 | 0

58. Secondary Outcome: Part D: Number of Participants With Positive Anti-TSR-042 Antibodies
Description: as for outcome 56
Time Frame: Up to 9.5 months
Population: Anti-drug Antibody Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab
Number analyzed (Participants) | 6
Participants | 0

59. Secondary Outcome: Part E: Number of Participants With Positive Anti-TSR-042 Antibodies
Description: as for outcome 56
Time Frame: Up to 4.4 months
Population: Anti-drug Antibody Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Part E: TSR-042 and Carboplatin-pemetrexed
Number analyzed (Participants) | 2
Participants | 0

60. Secondary Outcome: Part F: Number of Participants With Positive Anti-TSR-042 Antibodies
Description: as for outcome 56
Time Frame: Up to 3.5 months
Population: Anti-drug Antibody Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed
Number analyzed (Participants) | 1
Participants | NA — Data could not be calculated due to insufficient participant with data.

61. Secondary Outcome: Part F: Number of Participants With Positive Anti-TSR-022 Antibodies
Description: Serum samples were collected at indicated time points and tested for the presence of antibodies that bind to TSR-022. The presence of anti-TSR-022 antibodies were assessed using a tiered approach using electrochemiluminescence (that is, screening, confirmation, titer, and neutralizing antibody assay).
Time Frame: Up to 3.5 months
Population: Anti-drug Antibody Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed
Number analyzed (Participants) | 1
Participants | NA — Data could not be calculated due to insufficient participant with data.

62. Secondary Outcome: Part G: Number of Participants With Positive Anti-TSR-042 Antibodies
Description: Serum samples were planned to be collected at indicated time points and tested for the presence of antibodies that bind to TSR-042. The presence of anti-TSR-042 antibodies were planeed to be assessed using a tiered approach using electrochemiluminescence (that is, screening, confirmation, titer, and neutralizing antibody assay).
Time Frame: Up to 24 months
Population: Anti-drug Antibody Population. Data was not collected as no participants were enrolled in Part G.
Arm/Group | Main Study: Part G: TSR-042 and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

63. Secondary Outcome: Part H: Number of Participants With Positive Anti-TSR-042 Antibodies
Description: Serum samples were planned to be collected at indicated time points and tested for the presence of antibodies that bind to TSR-042. The presence of anti-TSR-042 antibodies were planned to be assessed using a tiered approach using electrochemiluminescence (that is, screening, confirmation, titer, and neutralizing antibody assay).
Time Frame: Up to 24 months
Population: Anti-drug Antibody Population. Data was not collected as no participants were enrolled in Part H.
Arm/Group | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

64. Secondary Outcome: Part H: Number of Participants With Positive Anti-TSR-022 Antibodies
Description: Serum samples were planned to be collected at indicated time points and tested for the presence of antibodies that bind to TSR-022. The presence of anti-TSR-022 antibodies were planned to be assessed using a tiered approach using electrochemiluminescence (that is, screening, confirmation, titer, and neutralizing antibody assay).
Time Frame: Up to 24 months
Population: Anti-drug Antibody Population. Data was not collected as no participants were enrolled in Part H.
Arm/Group | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

65. Secondary Outcome: Part I: Number of Participants With Positive Anti-TSR-042 Antibodies
Description: as for outcome 63
Time Frame: Up to 24 months
Population: Anti-drug Antibody Population. Data was not collected as no participants were enrolled in Part I.
Arm/Group | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel
Number analyzed (Participants) | 0

66. Secondary Outcome: Part I: Number of Participants With Positive Anti-TSR-022 Antibodies
Description: as for outcome 64
Time Frame: Up to 24 months
Population: Anti-drug Antibody Population. Data was not collected as no participants were enrolled in Part I.
Arm/Group | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel
Number analyzed (Participants) | 0

67. Secondary Outcome: Part A: Area Under the Plasma Concentration From Time Zero to t (AUC[0-t]) of Niraparib
Description: Blood samples were collected at indicated time points. Pharmacokinetic (PK) parameters of niraparib were calculated using non-compartmental methods. PK population consisted of all participants who received at least 1 dose of study treatment and had at least 1 PK sample.
Time Frame: Cycles 1 and 2: Pre-dose, 1, 2, 4, 6, 8 and 24 hours post-dose (each cycle was 21 days)
Population: PK Population. Only those participants with data available at the indicated time points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Hours*microgram per milliliter
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD
Number analyzed (Participants) | 15 | 6
Hours*microgram per milliliter
  Cycle 1, n=15,6 | 6.0430 (3.43261) | 7.8341 (4.76380)
  Cycle 2, n=10,3: number analyzed (Participants) | 10 | 3
  Cycle 2, n=10,3 | 14.9172 (9.82689) | 29.3024 (2.15129)

68. Secondary Outcome: Part A: AUC(0-t) of TSR-042
Description: Blood samples were collected at indicated time points. PK parameters of TSR-042 were calculated using non-compartmental methods.
Time Frame: Cycles 1 and 4: Pre-dose, 0.5, 2, 24, 96, 168, 336 and 504 hours post-dose; Cycles 5 and 11: Pre-dose, 0.5, 2, 24, 96, 168, 336, 504 and 1008 hours post-dose (each cycle was 21 days)
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Hours*microgram per milliliter
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD
Number analyzed (Participants) | 16 | 6
Hours*microgram per milliliter
  Cycle 1, n=16,6 | 26827.7703 (9811.74994) | 29420.8347 (9262.18751)
  Cycle 4, n=9,4: number analyzed (Participants) | 9 | 4
  Cycle 4, n=9,4 | 55408.3992 (21631.17124) | 29311.8182 (16546.73177)
  Cycle 5, n=8,1: number analyzed (Participants) | 8 | 1
  Cycle 5, n=8,1 | 137108.2574 (41494.15474) | 141328.9288 (NA) — Standard deviation could not be calculated for single participant.
  Cycle 11, n=5,0: number analyzed (Participants) | 5 | 0
  Cycle 11, n=5,0 | 139591.8834 (53844.12650) |

69. Secondary Outcome: Part B: AUC0-t of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 68
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Hours*microgram per milliliter
Arm/Group | Main Study: Part B: TSR-042 and Carboplatin-paclitaxel
Number analyzed (Participants) | 14
Hours*microgram per milliliter
  Cycle 1, n=14 | 28097.9846 (8440.50578)
  Cycle 4, n=10: number analyzed (Participants) | 10
  Cycle 4, n=10 | 54730.0053 (15857.69305)
  Cycle 5, n=9: number analyzed (Participants) | 9
  Cycle 5, n=9 | 124309.5455 (56505.10671)
  Cycle 11, n=6: number analyzed (Participants) | 6
  Cycle 11, n=6 | 117030.4081 (33852.45635)

70. Secondary Outcome: Part C: AUC0-t of Niraparib
Description: Blood samples were collected at indicated time points. PK parameters of niraparib were calculated using non-compartmental methods.
Time Frame: Cycles 1 and 2: Pre-dose, 1, 2, 4, 6, 8 and 24 hours post-dose (each cycle was 21 days)
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Hours*microgram per milliliter
Arm/Group | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab
Number analyzed (Participants) | 6 | 7
Hours*microgram per milliliter
  Cycle 1, n=6,7 | 3.4513 (1.23048) | 11.3601 (5.53524)
  Cycle 2, n=4,4: number analyzed (Participants) | 4 | 4
  Cycle 2, n=4,4 | 14.7473 (8.11715) | 24.9691 (17.50367)

71. Secondary Outcome: Part C: AUC0-t of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 68
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Hours*microgram per milliliter
Arm/Group | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab
Number analyzed (Participants) | 6 | 7
Hours*microgram per milliliter
  Cycle 1, n=6,7 | 29830.6542 (8143.36941) | 26311.1789 (4416.61957)
  Cycle 4, n=5,7: number analyzed (Participants) | 5 | 7
  Cycle 4, n=5,7 | 54268.1379 (14777.09545) | 49198.8237 (12507.66126)
  Cycle 5, n=5,6: number analyzed (Participants) | 5 | 6
  Cycle 5, n=5,6 | 137777.3188 (45794.21973) | 131281.9046 (36835.39730)
  Cycle 11, n=4,2: number analyzed (Participants) | 4 | 2
  Cycle 11, n=4,2 | 143070.3093 (74219.00272) | 119161.8795 (NA) — Standard deviation was not calculated as it is not statistically meaningful as there are only 2 participants.

72. Secondary Outcome: Part D: AUC0-t of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 68
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Hours*microgram per milliliter
Arm/Group | Main Study: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab
Number analyzed (Participants) | 6
Hours*microgram per milliliter
  Cycle 1, n=6 | 32819.5401 (9182.44511)
  Cycle 4, n=5: number analyzed (Participants) | 5
  Cycle 4, n=5 | 52409.0255 (11814.13244)
  Cycle 5, n=5: number analyzed (Participants) | 5
  Cycle 5, n=5 | 119847.0999 (27279.85524)
  Cycle 11, n=4: number analyzed (Participants) | 4
  Cycle 11, n=4 | 77794.6422 (38680.64753)

73. Secondary Outcome: Part E: AUC0-t of TSR-042
Description: as for outcome 68
Time Frame: Cycle 1: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose; Cycle 2: Pre-dose (each cycle was 21 days)
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Hours*microgram per milliliter
Arm/Group | Main Study: Part E: TSR-042 and Carboplatin-pemetrexed
Number analyzed (Participants) | 2
Hours*microgram per milliliter | NA (NA) — Data was not collected due to insufficient number of participants with data to calculate AUC0-t.

74. Secondary Outcome: Part F: AUC0-t of TSR-042
Description: as for outcome 68
Time Frame: Cycle 1: Pre-dose, 0.5, 1, 2, 3, 24, 48, 96, 168 and 336 hours post-dose; Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Hours*microgram per milliliter
Arm/Group | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed
Number analyzed (Participants) | 1
Hours*microgram per milliliter | NA (NA) — Data was not collected due to insufficient number of participants with data to calculate AUC0-t.

75. Secondary Outcome: Part F: AUC0-t of TSR-022
Description: Blood samples were collected at indicated time points. PK parameters of TSR-022 were calculated using non-compartmental methods.
Time Frame: as for outcome 74
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Hours*microgram per milliliter
Arm/Group | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed
Number analyzed (Participants) | 1
Hours*microgram per milliliter | NA (NA) — Data was not collected due to insufficient number of participants with data to calculate AUC0-t.

76. Secondary Outcome: Part G: AUC0-t of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycles 1 and 5: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose; Cycle 2: Pre-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part G.
Arm/Group | Main Study: Part G: TSR-042 and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

77. Secondary Outcome: Part H: AUC0-t of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: as for outcome 74
Population: PK Population. Data was not collected as no participants were enrolled in Part H.
Arm/Group | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

78. Secondary Outcome: Part H: AUC0-t of TSR-022
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: as for outcome 74
Population: PK Population. Data was not collected as no participants were enrolled in Part H.
Arm/Group | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

79. Secondary Outcome: Part I: AUC0-t of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: as for outcome 74
Population: PK Population. Data was not collected as no participants were enrolled in Part I.
Arm/Group | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel
Number analyzed (Participants) | 0

80. Secondary Outcome: Part I: AUC0-t of TSR-022
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: as for outcome 74
Population: PK Population. Data was not collected as no participants were enrolled in Part I.
Arm/Group | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel
Number analyzed (Participants) | 0

81. Secondary Outcome: Part A: Area Under the Plasma Concentration From Time Zero to Infinity (AUC[0-infinity]) of Niraparib
Description: as for outcome 70
Time Frame: Cycles 1 and 2: Pre-dose, 1, 2, 4, 6, 8 and 24 hours post-dose (each cycle was 21 days)
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD
Number analyzed (Participants) | 16 | 6
Hours*microgram per milliliter | NA (NA) — The terminal elimination phase could not be identified from the concentration-time profile over the study period; hence, AUC(0-infinity) could not be estimated. | NA (NA) — The terminal elimination phase could not be identified from the concentration-time profile over the study period; hence, AUC(0-infinity) could not be estimated.

82. Secondary Outcome: Part A: AUC(0-infinity) of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 68
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD
Number analyzed (Participants) | 16 | 6
Hours*microgram per milliliter | NA (NA) — The terminal elimination phase could not be identified from the concentration-time profile over the study period; hence, AUC(0-infinity) could not be estimated. | NA (NA) — The terminal elimination phase could not be identified from the concentration-time profile over the study period; hence, AUC(0-infinity) could not be estimated.

83. Secondary Outcome: Part B: AUC(0-infinity) of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 68
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Main Study: Part B: TSR-042 and Carboplatin-paclitaxel
Number analyzed (Participants) | 14
Hours*microgram per milliliter | NA (NA) — The terminal elimination phase could not be identified from the concentration-time profile over the study period; hence, AUC(0-infinity) could not be estimated.

84. Secondary Outcome: Part C: AUC(0-infinity) of Niraparib
Description: as for outcome 70
Time Frame: Cycles 1 and 2: Pre-dose, 1, 2, 4, 6, 8 and 24 hours post-dose (each cycle was 21 days)
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab
Number analyzed (Participants) | 6 | 7
Hours*microgram per milliliter | NA (NA) — The terminal elimination phase could not be identified from the concentration-time profile over the study period; hence, AUC(0-infinity) could not be estimated. | NA (NA) — The terminal elimination phase could not be identified from the concentration-time profile over the study period; hence, AUC(0-infinity) could not be estimated.

85. Secondary Outcome: Part C: AUC(0-infinity) of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 68
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab
Number analyzed (Participants) | 6 | 7
Hours*microgram per milliliter | NA (NA) — The terminal elimination phase could not be identified from the concentration-time profile over the study period; hence, AUC(0-infinity) could not be estimated. | NA (NA) — The terminal elimination phase could not be identified from the concentration-time profile over the study period; hence, AUC(0-infinity) could not be estimated.

86. Secondary Outcome: Part D: AUC(0-infinity) of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 68
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Main Study: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab
Number analyzed (Participants) | 6
Hours*microgram per milliliter | NA (NA) — The terminal elimination phase could not be identified from the concentration-time profile over the study period; hence, AUC(0-infinity) could not be estimated.

87. Secondary Outcome: Part E: AUC(0-infinity) of TSR-042
Description: as for outcome 68
Time Frame: Cycle 1: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose; Cycle 2: Pre-dose (each cycle was 21 days)
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Main Study: Part E: TSR-042 and Carboplatin-pemetrexed
Number analyzed (Participants) | 2
Hours*microgram per milliliter | NA (NA) — Data was not collected due to insufficient number of participants with data to calculate AUC(0-infinity).

88. Secondary Outcome: Part F: AUC(0-infinity) of TSR-042
Description: as for outcome 68
Time Frame: Cycle 1: Pre-dose, 0.5, 1, 2, 3, 24, 48, 96, 168, and 336 hours post-dose; Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed
Number analyzed (Participants) | 1
Hours*microgram per milliliter | NA (NA) — Data was not collected due to insufficient number of participants with data to calculate AUC(0-infinity).

89. Secondary Outcome: Part F: AUC(0-infinity) of TSR-022
Description: as for outcome 75
Time Frame: Cycle 1: Pre-dose, 0.5, 1, 2, 3, 24, 48, 96, 168 and 336 hours post-dose; Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 48, 96, 168 and 336 hours post-dose (each cycle was 21 days)
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed
Number analyzed (Participants) | 1
Hours*microgram per milliliter | NA (NA) — Data was not collected due to insufficient number of participants with data to calculate AUC(0-infinity).

90. Secondary Outcome: Part G: AUC(0-infinity) of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycles 1 and 5: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose; Cycle 2: Pre-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part G.
Arm/Group | Main Study: Part G: TSR-042 and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

91. Secondary Outcome: Part H: AUC(0-infinity) of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 1: Pre-dose, 0.5, 1, 2, 3, 24, 48, 96, 168 and 336 hours post-dose; Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part H.
Arm/Group | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

92. Secondary Outcome: Part H: AUC(0-infinity) of TSR-022
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: as for outcome 91
Population: PK Population. Data was not collected as no participants were enrolled in Part H.
Arm/Group | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

93. Secondary Outcome: Part I: AUC(0-infinity) of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: as for outcome 74
Population: PK Population. Data was not collected as no participants were enrolled in Part I.
Arm/Group | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel
Number analyzed (Participants) | 0

94. Secondary Outcome: Part I: AUC(0-infinity) of TSR-022
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: as for outcome 74
Population: PK Population. Data was not collected as no participants were enrolled in Part I.
Arm/Group | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel
Number analyzed (Participants) | 0

95. Secondary Outcome: Part A: Observed Concentration at the End of the Dosing Interval (Ctau) of Niraparib
Description: as for outcome 70
Time Frame: Cycle 1: Pre-dose, 1, 2, 4, 6, 8 and 24 hours post-dose (each cycle was 21 days)
Population: PK Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD
Number analyzed (Participants) | 15 | 6
Microgram per milliliter | 0.191953 (0.1309536) | 0.342333 (0.3301392)

96. Secondary Outcome: Part A: Ctau of TSR-042
Description: as for outcome 68
Time Frame: Cycle 1: Pre-dose, 0.5, 2, 24, 96, 168, 336 and 504 hours post-dose (each cycle was 21 days)
Population: PK Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD
Number analyzed (Participants) | 9 | 4
Microgram per milliliter | 33.6000 (12.25194) | 29.8000 (10.32570)

97. Secondary Outcome: Part B: Ctau of TSR-042
Description: as for outcome 68
Time Frame: Cycle 1: Pre-dose, 0.5, 2, 24, 96, 168, 336 and 504 hours post-dose (each cycle was 21 days)
Population: PK Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part B: TSR-042 and Carboplatin-paclitaxel
Number analyzed (Participants) | 9
Microgram per milliliter | 33.9778 (9.89846)

98. Secondary Outcome: Part C: Ctau of Niraparib
Description: as for outcome 70
Time Frame: Cycle 1: Pre-dose, 1, 2, 4, 6, 8 and 24 hours post-dose (each cycle was 21 days)
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab
Number analyzed (Participants) | 6 | 7
Microgram per milliliter | 0.161233 (0.1072328) | 0.478714 (0.4197538)

99. Secondary Outcome: Part C: Ctau of TSR-042
Description: as for outcome 68
Time Frame: Cycle 1: Pre-dose, 0.5, 2, 24, 96, 168, 336 and 504 hours post-dose (each cycle was 21 days)
Population: PK Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab
Number analyzed (Participants) | 4 | 4
Microgram per milliliter | 37.2750 (16.78102) | 28.7500 (9.47505)

100. Secondary Outcome: Part D: Ctau of TSR-042
Description: as for outcome 68
Time Frame: Cycle 1: Pre-dose, 0.5, 2, 24, 96, 168, 336 and 504 hours post-dose (each cycle was 21 days)
Population: PK Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab
Number analyzed (Participants) | 4
Microgram per milliliter | 36.5250 (12.29834)

101. Secondary Outcome: Part E: Ctau of TSR-042
Description: as for outcome 68
Time Frame: Cycle 1: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part E: TSR-042 and Carboplatin-pemetrexed
Number analyzed (Participants) | 2
Microgram per milliliter | NA (NA) — Data was not collected due to insufficient number of participants with data to calculate Ctau.

102. Secondary Outcome: Part F: Ctau of TSR-042
Description: as for outcome 68
Time Frame: Cycle 1: Pre-dose, 0.5, 1, 2, 3, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed
Number analyzed (Participants) | 1
Microgram per milliliter | NA (NA) — Data was not collected due to insufficient number of participants with data to calculate Ctau.

103. Secondary Outcome: Part F: Ctau of TSR-022
Description: as for outcome 75
Time Frame: Cycle 1: Pre-dose, 0.5, 1, 2, 3, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed
Number analyzed (Participants) | 1
Microgram per milliliter | NA (NA) — Data was not collected due to insufficient number of participants with data to calculate Ctau.

104. Secondary Outcome: Part G: Ctau of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 1: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part G.
Arm/Group | Main Study: Part G: TSR-042 and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

105. Secondary Outcome: Part H: Ctau of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 1: Pre-dose, 0.5, 1, 2, 3, 24, 48, 96, 168 and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part H.
Arm/Group | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

106. Secondary Outcome: Part H: Ctau of TSR-022
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 1: Pre-dose, 0.5, 1, 2, 3, 24, 48, 96, 168 and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part H.
Arm/Group | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

107. Secondary Outcome: Part I: Ctau of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 1: Pre-dose, 0.5, 1, 2, 3, 24, 48, 96, 168 and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part I.
Arm/Group | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel
Number analyzed (Participants) | 0

108. Secondary Outcome: Part I: Ctau of TSR-022
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 1: Pre-dose, 0.5, 1, 2, 3, 24, 48, 96, 168 and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part I.
Arm/Group | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel
Number analyzed (Participants) | 0

109. Secondary Outcome: Part A: Maximum Observed Plasma (Cmax) of Niraparib
Description: as for outcome 70
Time Frame: Cycle 1: Pre-dose, 1, 2, 4, 6, 8 and 24 hours post-dose (each cycle was 21 days)
Population: PK Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD
Number analyzed (Participants) | 15 | 6
Microgram per milliliter | 0.460600 (0.2401100) | 0.625667 (0.4547692)

110. Secondary Outcome: Part A: Cmax of TSR-042
Description: as for outcome 68
Time Frame: Cycle 1: Pre-dose, 0.5, 2, 24, 96, 168, 336 and 504 hours post-dose (each cycle was 21 days)
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD
Number analyzed (Participants) | 16 | 6
Microgram per milliliter | 158.6875 (27.70251) | 138.9167 (37.87930)

111. Secondary Outcome: Part B: Cmax of TSR-042
Description: as for outcome 68
Time Frame: Cycle 1: Pre-dose, 0.5, 2, 24, 96, 168, 336 and 504 hours post-dose (each cycle was 21 days)
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part B: TSR-042 and Carboplatin-paclitaxel
Number analyzed (Participants) | 14
Microgram per milliliter | 148.2000 (31.27948)

112. Secondary Outcome: Part C: Cmax of Niraparib
Description: as for outcome 70
Time Frame: Cycle 1: Pre-dose, 1, 2, 4, 6, 8 and 24 hours post-dose (each cycle was 21 days)
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab
Number analyzed (Participants) | 6 | 7
Microgram per milliliter | 0.243667 (0.0889936) | 0.891571 (0.4638897)

113. Secondary Outcome: Part C: Cmax of TSR-042
Description: as for outcome 68
Time Frame: Cycle 1: Pre-dose, 0.5, 2, 24, 96, 168, 336 and 504 hours post-dose (each cycle was 21 days)
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab
Number analyzed (Participants) | 6 | 7
Microgram per milliliter | 138.6667 (24.14677) | 158.4857 (48.36788)

114. Secondary Outcome: Part D: Cmax of TSR-042
Description: as for outcome 68
Time Frame: Cycle 1: Pre-dose, 0.5, 2, 24, 96, 168, 336 and 504 hours post-dose (each cycle was 21 days)
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab
Number analyzed (Participants) | 6
Microgram per milliliter | 188.5000 (36.04858)

115. Secondary Outcome: Part E: Cmax of TSR-042
Description: as for outcome 68
Time Frame: Cycle 1: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part E: TSR-042 and Carboplatin-pemetrexed
Number analyzed (Participants) | 2
Microgram per milliliter | NA (NA) — Data was not collected due to insufficient number of participants with data to calculate Cmax.

116. Secondary Outcome: Part F: Cmax of TSR-042
Description: as for outcome 68
Time Frame: Cycle 1: Pre-dose, 0.5, 1, 2, 3, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed
Number analyzed (Participants) | 1
Microgram per milliliter | NA (NA) — Data was not collected due to insufficient number of participants with data to calculate Cmax.

117. Secondary Outcome: Part F: Cmax of TSR-022
Description: as for outcome 75
Time Frame: Cycle 1: Pre-dose, 0.5, 1, 2, 3, 24, 48, 96, 168 and 336 hours post-dose (each cycle was 21 days)
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed
Number analyzed (Participants) | 1
Microgram per milliliter | NA (NA) — Data was not collected due to insufficient number of participants with data to calculate Cmax.

118. Secondary Outcome: Part G: Cmax of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 1: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part G.
Arm/Group | Main Study: Part G: TSR-042 and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

119. Secondary Outcome: Part H: Cmax of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 1: Pre-dose, 0.5, 1, 2, 3, 24, 48, 96, 168 and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part H.
Arm/Group | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

120. Secondary Outcome: Part H: Cmax of TSR-022
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 1: Pre-dose, 0.5, 1, 2, 3, 24, 48, 96, 168 and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part H.
Arm/Group | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

121. Secondary Outcome: Part I: Cmax of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 1: Pre-dose, 0.5, 1, 2, 3, 24, 48, 96, 168 and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part I.
Arm/Group | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel
Number analyzed (Participants) | 0

122. Secondary Outcome: Part I: Cmax of TSR-022
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 1: Pre-dose, 0.5, 1, 2, 3, 24, 48, 96, 168 and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part I.
Arm/Group | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel
Number analyzed (Participants) | 0

123. Secondary Outcome: Part A: Clearance After Oral Administration (CL/F) of Niraparib
Description: as for outcome 70
Time Frame: Cycles 1 and 2: Pre-dose, 1, 2, 4, 6, 8 and 24 hours post-dose (each cycle was 21 days)
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Liter per hour
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD
Number analyzed (Participants) | 8 | 2
Liter per hour
  Cycle 1, n=1,0: number analyzed (Participants) | 1 | 0
  Cycle 1, n=1,0 | 28.5638 (NA) — Standard deviation could not be calculated for single participant. |
  Cycle 2, n=8,2 | 16.6295 (8.70836) | 10.2833 (NA) — Standard deviation was not calculated as it is not statistically meaningful as there are only 2 participants.

124. Secondary Outcome: Part A: Clearance After Intravenous Administration (CL) of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 68
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Liter per hour
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD
Number analyzed (Participants) | 8 | 2
Liter per hour
  Cycle 1, n=0,0: number analyzed (Participants) | 0 | 0
  Cycle 4, n=7,2: number analyzed (Participants) | 7 | 2
  Cycle 4, n=7,2 | 0.0090 (0.00220) | 0.0110 (NA) — Standard deviation was not calculated as it is not statistically meaningful as there are only 2 participants.
  Cycle 5, n=8,1: number analyzed (Participants) | 8 | 1
  Cycle 5, n=8,1 | 0.0081 (0.00238) | 0.0071 (NA) — Standard deviation could not be calculated for single participant.
  Cycle 11, n=4,0: number analyzed (Participants) | 4 | 0
  Cycle 11, n=4,0 | 0.0072 (0.00217) |

125. Secondary Outcome: Part B: CL of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 68
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Liter per hour
Arm/Group | Main Study: Part B: TSR-042 and Carboplatin-paclitaxel
Number analyzed (Participants) | 10
Liter per hour
  Cycle 1, n=0: number analyzed (Participants) | 0
  Cycle 4, n=10 | 0.0098 (0.00292)
  Cycle 5, n=8: number analyzed (Participants) | 8
  Cycle 5, n=8 | 0.0082 (0.00242)
  Cycle 11, n=6: number analyzed (Participants) | 6
  Cycle 11, n=6 | 0.0092 (0.00296)

126. Secondary Outcome: Part C: CL/F of Niraparib
Description: as for outcome 70
Time Frame: Cycles 1 and 2: Pre-dose, 1, 2, 4, 6, 8 and 24 hours post-dose (each cycle was 21 days)
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Liter per hour
Arm/Group | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab
Number analyzed (Participants) | 2 | 4
Liter per hour
  Cycle 1, n=0,0: number analyzed (Participants) | 0 | 0
  Cycle 2, n=2,4 | 10.3777 (NA) — Standard deviation was not calculated as it is not statistically meaningful as there are only 2 participants. | 14.4947 (8.40967)

127. Secondary Outcome: Part C: CL of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 68
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Liter per hour
Arm/Group | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab
Number analyzed (Participants) | 5 | 6
Liter per hour
  Cycle 1, n=0,0: number analyzed (Participants) | 0 | 0
  Cycle 4, n=5,5: number analyzed (Participants) | 5 | 5
  Cycle 4, n=5,5 | 0.0100 (0.00441) | 0.0104 (0.00268)
  Cycle 5, n=5,6 | 0.0082 (0.00370) | 0.0082 (0.00273)
  Cycle 11, n=4,2: number analyzed (Participants) | 4 | 2
  Cycle 11, n=4,2 | 0.0079 (0.00391) | 0.0086 (NA) — Standard deviation was not calculated as it is not statistically meaningful as there are only 2 participants.

128. Secondary Outcome: Part D: CL of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 68
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Liter per hour
Arm/Group | Main Study: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab
Number analyzed (Participants) | 5
Liter per hour
  Cycle 1, n=0: number analyzed (Participants) | 0
  Cycle 4, n=5 | 0.0102 (0.00210)
  Cycle 5, n=5 | 0.0087 (0.00169)
  Cycle 11, n=3: number analyzed (Participants) | 3
  Cycle 11, n=3 | 0.0104 (0.00100)

129. Secondary Outcome: Part E: CL of TSR-042
Description: as for outcome 68
Time Frame: Cycle 1: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose; Cycle 2: Pre-dose (each cycle was 21 days)
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Liter per hour
Arm/Group | Main Study: Part E: TSR-042 and Carboplatin-pemetrexed
Number analyzed (Participants) | 2
Liter per hour | NA (NA) — Data was not collected due to insufficient number of participants with data to calculate CL.

130. Secondary Outcome: Part F: CL of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 88
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Liter per hour
Arm/Group | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed
Number analyzed (Participants) | 1
Liter per hour | NA (NA) — Data was not collected due to insufficient number of participants with data to calculate CL.

131. Secondary Outcome: Part F: CL of TSR-022
Description: as for outcome 75
Time Frame: as for outcome 88
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Liter per hour
Arm/Group | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed
Number analyzed (Participants) | 1
Liter per hour | NA (NA) — Data was not collected due to insufficient number of participants with data to calculate CL.

132. Secondary Outcome: Part G: CL of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycles 1 and 5: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose; Cycle 2: Pre-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part G.
Arm/Group | Main Study: Part G: TSR-042 and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

133. Secondary Outcome: Part H: CL of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: as for outcome 91
Population: PK Population. Data was not collected as no participants were enrolled in Part H.
Arm/Group | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

134. Secondary Outcome: Part H: CL of TSR-022
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: as for outcome 91
Population: PK Population. Data was not collected as no participants were enrolled in Part H.
Arm/Group | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

135. Secondary Outcome: Part I: CL of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: as for outcome 74
Population: PK Population. Data was not collected as no participants were enrolled in Part I.
Arm/Group | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel
Number analyzed (Participants) | 0

136. Secondary Outcome: Part I: CL of TSR-022
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: as for outcome 74
Population: PK Population. Data was not collected as no participants were enrolled in Part I.
Arm/Group | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel
Number analyzed (Participants) | 0

137. Secondary Outcome: Part A: Volume of Distribution After Oral Administration (Vz/F) of Niraparib
Description: as for outcome 70
Time Frame: Cycles 1 and 2: Pre-dose, 1, 2, 4, 6, 8 and 24 hours post-dose (each cycle was 21 days)
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD
Number analyzed (Participants) | 8 | 2
Liter
  Cycle 1, n=1,0: number analyzed (Participants) | 1 | 0
  Cycle 1, n=1,0 | 380.1478 (NA) — Standard deviation could not be calculated for single participant. |
  Cycle 2, n=8,2 | 716.1418 (554.80278) | 487.8826 (NA) — Standard deviation was not calculated as it is not statistically meaningful as there are only 2 participants.

138. Secondary Outcome: Part A: Volume of Distribution After Intravenous Administration (Vz) of of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 68
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD
Number analyzed (Participants) | 8 | 2
Liter
  Cycle 1, n=0,0: number analyzed (Participants) | 0 | 0
  Cycle 4, n=5,2: number analyzed (Participants) | 5 | 2
  Cycle 4, n=5,2 | 5.6925 (1.46062) | 10.3984 (NA) — Standard deviation was not calculated as it is not statistically meaningful as there are only 2 participants.
  Cycle 5, n=8,1: number analyzed (Participants) | 8 | 1
  Cycle 5, n=8,1 | 6.8811 (1.70545) | 6.3070 (NA) — Standard deviation could not be calculated for single participant.
  Cycle 11, n=4,0: number analyzed (Participants) | 4 | 0
  Cycle 11, n=4,0 | 7.4795 (0.90952) |

139. Secondary Outcome: Part B: Vz of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 68
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Main Study: Part B: TSR-042 and Carboplatin-paclitaxel
Number analyzed (Participants) | 10
Liter
  Cycle 1, n=0: number analyzed (Participants) | 0
  Cycle 4, n=10 | 5.3661 (2.01321)
  Cycle 5, n=8: number analyzed (Participants) | 8
  Cycle 5, n=8 | 7.2627 (2.43311)
  Cycle 11, n=6: number analyzed (Participants) | 6
  Cycle 11, n=6 | 8.0529 (3.64454)

140. Secondary Outcome: Part C: Vz/F of Niraparib
Description: as for outcome 70
Time Frame: Cycles 1 and 2: Pre-dose, 1, 2, 4, 6, 8 and 24 hours post-dose (each cycle was 21 days)
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab
Number analyzed (Participants) | 2 | 2
Liter
  Cycle 1, n=0,0: number analyzed (Participants) | 0 | 0
  Cycle 2, n=2,2 | 551.4003 (NA) — Standard deviation was not calculated as it is not statistically meaningful as there are only 2 participants. | 559.3634 (NA) — Standard deviation was not calculated as it is not statistically meaningful as there are only 2 participants.

141. Secondary Outcome: Part C: Vz of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 68
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab
Number analyzed (Participants) | 5 | 6
Liter
  Cycle 1, n=0,0: number analyzed (Participants) | 0 | 0
  Cycle 4, n=5,5: number analyzed (Participants) | 5 | 5
  Cycle 4, n=5,5 | 6.6462 (2.66825) | 5.8922 (2.93257)
  Cycle 5, n=4,6: number analyzed (Participants) | 4 | 6
  Cycle 5, n=4,6 | 6.1698 (1.73272) | 5.2066 (1.07206)
  Cycle 11, n=4,2: number analyzed (Participants) | 4 | 2
  Cycle 11, n=4,2 | 9.6347 (4.05466) | 8.5098 (NA) — Standard deviation was not calculated as it is not statistically meaningful as there are only 2 participants.

142. Secondary Outcome: Part D: Vz of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 68
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Main Study: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab
Number analyzed (Participants) | 5
Liter
  Cycle 1, n=0: number analyzed (Participants) | 0
  Cycle 4, n=5 | 5.4955 (1.89543)
  Cycle 5, n=5 | 6.1542 (1.57345)
  Cycle 11, n=3: number analyzed (Participants) | 3
  Cycle 11, n=3 | 9.8356 (0.99107)

143. Secondary Outcome: Part E: Vz of TSR-042
Description: as for outcome 68
Time Frame: Cycle 1: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose; Cycle 2: Pre-dose (each cycle was 21 days)
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Main Study: Part E: TSR-042 and Carboplatin-pemetrexed
Number analyzed (Participants) | 2
Liter | NA (NA) — Data was not collected due to insufficient number of participants with data to calculate Vz.

144. Secondary Outcome: Part F: Vz of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 88
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed
Number analyzed (Participants) | 1
Liter | NA (NA) — Data was not collected due to insufficient number of participants with data to calculate Vz.

145. Secondary Outcome: Part F: Vz of TSR-022
Description: as for outcome 75
Time Frame: as for outcome 88
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed
Number analyzed (Participants) | 1
Liter | NA (NA) — Data was not collected due to insufficient number of participants with data to calculate Vz.

146. Secondary Outcome: Part G: Vz of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycles 1 and 5: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose; Cycle 2: Pre-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part G.
Arm/Group | Main Study: Part G: TSR-042 and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

147. Secondary Outcome: Part H: Vz of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: as for outcome 91
Population: PK Population. Data was not collected as no participants were enrolled in Part H.
Arm/Group | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

148. Secondary Outcome: Part H: Vz of TSR-022
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: as for outcome 91
Population: PK Population. Data was not collected as no participants were enrolled in Part H.
Arm/Group | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

149. Secondary Outcome: Part I: Vz of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: as for outcome 74
Population: PK Population. Data was not collected as no participants were enrolled in Part I.
Arm/Group | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel
Number analyzed (Participants) | 0

150. Secondary Outcome: Part I: Vz of TSR-022
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: as for outcome 74
Population: PK Population. Data was not collected as no participants were enrolled in Part I.
Arm/Group | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel
Number analyzed (Participants) | 0

151. Secondary Outcome: Part A: AUC at Steady State (AUCss) of Niraparib
Description: as for outcome 70
Time Frame: Cycle 2: Pre-dose, 1, 2, 4, 6, 8 and 24 hours post-dose (each cycle was 21 days)
Population: PK Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Hours*microgram per milliliter
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD
Number analyzed (Participants) | 8 | 2
Hours*microgram per milliliter | 16.3481 (10.63803) | 29.4312 (NA) — Standard deviation was not calculated as it is not statistically meaningful as there are only 2 participants.

152. Secondary Outcome: Part A: AUCss of TSR-042
Description: as for outcome 68
Time Frame: Cycle 4: Pre-dose, 0.5, 2, 24, 96, 168, 336 and 504 hours post-dose; Cycles 5 and 11: Pre-dose, 0.5, 2, 24, 96, 168, 336, 504 and 1008 hours post-dose (each cycle was 21 days)
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Hours*microgram per milliliter
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD
Number analyzed (Participants) | 8 | 3
Hours*microgram per milliliter
  Cycle 4, n=7,2: number analyzed (Participants) | 7 | 2
  Cycle 4, n=7,2 | 58598.5076 (15328.61731) | 46122.3924 (NA) — Standard deviation was not calculated as it is not statistically meaningful as there are only 2 participants.
  Cycle 5, n=8,1: number analyzed (Participants) | 8 | 1
  Cycle 5, n=8,1 | 135171.2753 (43806.32512) | 141306.3782 (NA) — Standard deviation could not be calculated for single participant.
  Cycle 11, n=4,0: number analyzed (Participants) | 4 | 0
  Cycle 11, n=4,0 | 151575.3645 (55194.65972) |

153. Secondary Outcome: Part B: AUCss of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 152
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Hours*microgram per milliliter
Arm/Group | Main Study: Part B: TSR-042 and Carboplatin-paclitaxel
Number analyzed (Participants) | 10
Hours*microgram per milliliter
  Cycle 4, n=10 | 55073.0926 (15304.21896)
  Cycle 5, n=8: number analyzed (Participants) | 8
  Cycle 5, n=8 | 130694.9752 (33923.75772)
  Cycle 11, n=6: number analyzed (Participants) | 6
  Cycle 11, n=6 | 117033.3612 (33727.51653)

154. Secondary Outcome: Part C: AUCss of Niraparib
Description: as for outcome 70
Time Frame: Cycle 2: Pre-dose, 1, 2, 4, 6, 8 and 24 hours post-dose (each cycle was 21 days)
Population: PK Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Hours*microgram per milliliter
Arm/Group | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab
Number analyzed (Participants) | 2 | 4
Hours*microgram per milliliter | 21.4926 (NA) — Standard deviation was not calculated as it is not statistically meaningful as there are only 2 participants. | 26.5006 (14.61077)

155. Secondary Outcome: Part C: AUCss of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 152
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Hours*microgram per milliliter
Arm/Group | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab
Number analyzed (Participants) | 5 | 6
Hours*microgram per milliliter
  Cycle 4, n=5,5: number analyzed (Participants) | 5 | 5
  Cycle 4, n=5,5 | 55974.4268 (16738.05254) | 50924.1510 (13339.28085)
  Cycle 5, n=5,6 | 137399.5881 (45511.62023) | 131288.0291 (36816.18787)
  Cycle 11, n=4,2: number analyzed (Participants) | 4 | 2
  Cycle 11, n=4,2 | 147907.5379 (60795.87607) | 119189.5905 (NA) — Standard deviation was not calculated as it is not statistically meaningful as there are only 2 participants.

156. Secondary Outcome: Part D: AUCss of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 152
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Hours*microgram per milliliter
Arm/Group | Main Study: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab
Number analyzed (Participants) | 5
Hours*microgram per milliliter
  Cycle 4, n=5 | 51140.4410 (12597.07380)
  Cycle 5, n=5 | 118845.3928 (27874.98871)
  Cycle 11, n=3: number analyzed (Participants) | 3
  Cycle 11, n=3 | 96800.1534 (8871.32089)

157. Secondary Outcome: Part E: AUCss of TSR-042
Description: as for outcome 68
Time Frame: Cycle 2: Pre-dose (each cycle was 21 days)
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Hours*microgram per milliliter
Arm/Group | Main Study: Part E: TSR-042 and Carboplatin-pemetrexed
Number analyzed (Participants) | 2
Hours*microgram per milliliter | NA (NA) — Data was not collected due to insufficient number of participants with data to calculate AUCss.

158. Secondary Outcome: Part F: AUCss of TSR-042
Description: as for outcome 68
Time Frame: Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Hours*microgram per milliliter
Arm/Group | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed
Number analyzed (Participants) | 1
Hours*microgram per milliliter | NA (NA) — Data was not collected due to insufficient number of participants with data to calculate AUCss.

159. Secondary Outcome: Part F: AUCss of TSR-022
Description: as for outcome 75
Time Frame: Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Hours*microgram per milliliter
Arm/Group | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed
Number analyzed (Participants) | 1
Hours*microgram per milliliter | NA (NA) — Data was not collected due to insufficient number of participants with data to calculate AUCss.

160. Secondary Outcome: Part G: AUCss of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part G.
Arm/Group | Main Study: Part G: TSR-042 and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

161. Secondary Outcome: Part H: AUCss of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part H.
Arm/Group | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

162. Secondary Outcome: Part H: AUCss of TSR-022
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part H.
Arm/Group | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

163. Secondary Outcome: Part I: AUCss of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part I.
Arm/Group | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel
Number analyzed (Participants) | 0

164. Secondary Outcome: Part I: AUCss of TSR-022
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part I.
Arm/Group | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel
Number analyzed (Participants) | 0

165. Secondary Outcome: Part A: Ctau at Steady State (Ctau,ss) of Niraparib
Description: as for outcome 70
Time Frame: Cycle 2: Pre-dose, 1, 2, 4, 6, 8 and 24 hours post-dose; Cycles 5 and 11: Pre-dose, 2 hours post-dose (each cycle was 21 days)
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD
Number analyzed (Participants) | 11 | 6
Microgram per milliliter
  Cycle 2, n=11,6 | 0.507900 (0.3937657) | 0.622000 (0.4523848)
  Cycle 5, n=0,0: number analyzed (Participants) | 0 | 0
  Cycle 11, n=0,0: number analyzed (Participants) | 0 | 0

166. Secondary Outcome: Part A: Ctau,ss of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 152
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD
Number analyzed (Participants) | 8 | 1
Microgram per milliliter
  Cycle 4, n=8,1 | 77.3625 (28.55145) | 63.3000 (NA) — Standard deviation could not be calculated for single participant.
  Cycle 5, n=8,1 | 68.5500 (34.63879) | 71.2000 (NA) — Standard deviation could not be calculated for single participant.
  Cycle 11, n=4,0: number analyzed (Participants) | 4 | 0
  Cycle 11, n=4,0 | 93.8000 (47.28939) |

167. Secondary Outcome: Part B: Ctau,ss of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 152
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part B: TSR-042 and Carboplatin-paclitaxel
Number analyzed (Participants) | 9
Microgram per milliliter
  Cycle 4, n=9 | 67.2444 (24.15130)
  Cycle 5, n=8: number analyzed (Participants) | 8
  Cycle 5, n=8 | 59.3000 (16.75913)
  Cycle 11, n=6: number analyzed (Participants) | 6
  Cycle 11, n=6 | 57.4833 (20.98136)

168. Secondary Outcome: Part C: Ctau,ss of Niraparib
Description: as for outcome 70
Time Frame: as for outcome 165
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab
Number analyzed (Participants) | 5 | 4
Microgram per milliliter
  Cycle 2, n=5,4 | 0.484000 (0.3511339) | 1.094250 (0.7660576)
  Cycle 5, n=0,0: number analyzed (Participants) | 0 | 0
  Cycle 11, n=0,0: number analyzed (Participants) | 0 | 0

169. Secondary Outcome: Part C: Ctau,ss of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 152
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab
Number analyzed (Participants) | 5 | 6
Microgram per milliliter
  Cycle 4, n=4,6: number analyzed (Participants) | 4 | 6
  Cycle 4, n=4,6 | 70.4250 (34.00896) | 64.2667 (23.55315)
  Cycle 5, n=5,6 | 82.9800 (43.98252) | 53.1500 (24.80538)
  Cycle 11, n=3,2: number analyzed (Participants) | 3 | 2
  Cycle 11, n=3,2 | 105.4667 (22.28909) | 60.9500 (NA) — Standard deviation was not calculated as it is not statistically meaningful as there are only 2 participants.

170. Secondary Outcome: Part D: Ctau,ss of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 152
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab
Number analyzed (Participants) | 5
Microgram per milliliter
  Cycle 4, n=5 | 53.5200 (13.87271)
  Cycle 5, n=5 | 48.0800 (23.95343)
  Cycle 11, n=3: number analyzed (Participants) | 3
  Cycle 11, n=3 | 43.3000 (4.80729)

171. Secondary Outcome: Part E: Ctau,ss of TSR-042
Description: as for outcome 68
Time Frame: Cycle 2: Pre-dose (each cycle was 21 days)
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part E: TSR-042 and Carboplatin-pemetrexed
Number analyzed (Participants) | 2
Microgram per milliliter | NA (NA) — Data was not collected due to insufficient number of participants with data to calculate Ctau,ss.

172. Secondary Outcome: Part F: Ctau,ss of TSR-042
Description: as for outcome 68
Time Frame: Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed
Number analyzed (Participants) | 1
Microgram per milliliter | NA (NA) — Data was not collected due to insufficient number of participants with data to calculate Ctau,ss.

173. Secondary Outcome: Part F: Ctau,ss of TSR-022
Description: as for outcome 75
Time Frame: Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed
Number analyzed (Participants) | 1
Microgram per milliliter | NA (NA) — Data was not collected due to insufficient number of participants with data to calculate Ctau,ss.

174. Secondary Outcome: Part G: Ctau,ss of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part G.
Arm/Group | Main Study: Part G: TSR-042 and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

175. Secondary Outcome: Part H: Ctau,ss of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part H.
Arm/Group | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

176. Secondary Outcome: Part H: Ctau,ss of TSR-022
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part H.
Arm/Group | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

177. Secondary Outcome: Part I: Ctau,ss of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part I.
Arm/Group | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel
Number analyzed (Participants) | 0

178. Secondary Outcome: Part I: Ctau,ss of TSR-022
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part I.
Arm/Group | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel
Number analyzed (Participants) | 0

179. Secondary Outcome: Part A: Cmax at Steady State (Cmax,ss) of Niraparib
Description: as for outcome 70
Time Frame: as for outcome 165
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD
Number analyzed (Participants) | 10 | 3
Microgram per milliliter
  Cycle 2, n=10,3 | 0.925900 (0.6661597) | 1.706667 (0.0838650)
  Cycle 5, n=7,0: number analyzed (Participants) | 7 | 0
  Cycle 5, n=7,0 | 0.839071 (0.6183628) |
  Cycle 11, n=2,0: number analyzed (Participants) | 2 | 0
  Cycle 11, n=2,0 | 0.768000 (NA) — Standard deviation was not calculated as it is not statistically meaningful as there are only 2 participants. |

180. Secondary Outcome: Part A: Cmax,ss of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 152
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD
Number analyzed (Participants) | 9 | 4
Microgram per milliliter
  Cycle 4, n=9,4 | 222.5556 (51.37633) | 178.5000 (26.18524)
  Cycle 5, n=8,1: number analyzed (Participants) | 8 | 1
  Cycle 5, n=8,1 | 393.8750 (100.81729) | 319.0000 (NA) — Standard deviation could not be calculated for single participant.
  Cycle 11, n=5,0: number analyzed (Participants) | 5 | 0
  Cycle 11, n=5,0 | 405.4000 (103.69812) |

181. Secondary Outcome: Part B: Cmax,ss of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 152
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part B: TSR-042 and Carboplatin-paclitaxel
Number analyzed (Participants) | 10
Microgram per milliliter
  Cycle 4, n=10 | 225.8000 (51.71460)
  Cycle 5, n=9: number analyzed (Participants) | 9
  Cycle 5, n=9 | 421.1111 (114.84603)
  Cycle 11, n=6: number analyzed (Participants) | 6
  Cycle 11, n=6 | 446.6667 (160.53868)

182. Secondary Outcome: Part C: Cmax,ss of Niraparib
Description: as for outcome 70
Time Frame: as for outcome 165
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab
Number analyzed (Participants) | 4 | 4
Microgram per milliliter
  Cycle 2, n=4,4 | 0.854500 (0.3934637) | 1.404750 (0.6642366)
  Cycle 5, n=4,3: number analyzed (Participants) | 4 | 3
  Cycle 5, n=4,3 | 0.709750 (0.2693788) | 1.073667 (0.5474124)
  Cycle 11, n=3,1: number analyzed (Participants) | 3 | 1
  Cycle 11, n=3,1 | 0.468333 (0.1418955) | 0.638000 (NA) — Standard deviation could not be calculated for single participant.

183. Secondary Outcome: Part C: Cmax,ss of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 152
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab
Number analyzed (Participants) | 5 | 7
Microgram per milliliter
  Cycle 4, n=5,7 | 234.4000 (31.76948) | 227.1429 (42.65923)
  Cycle 5, n=5,6: number analyzed (Participants) | 5 | 6
  Cycle 5, n=5,6 | 325.2000 (73.90332) | 417.3333 (139.40397)
  Cycle 11, n=4,2: number analyzed (Participants) | 4 | 2
  Cycle 11, n=4,2 | 349.7500 (111.53886) | 321.0000 (NA) — Standard deviation was not calculated as it is not statistically meaningful as there are only 2 participants.

184. Secondary Outcome: Part D: Cmax,ss of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 152
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab
Number analyzed (Participants) | 5
Microgram per milliliter
  Cycle 4, n=5 | 256.8000 (76.90709)
  Cycle 5, n=5 | 416.0000 (89.43433)
  Cycle 11, n=4: number analyzed (Participants) | 4
  Cycle 11, n=4 | 429.7500 (72.86231)

185. Secondary Outcome: Part E: Cmax,ss of TSR-042
Description: as for outcome 68
Time Frame: Cycle 2: Pre-dose (each cycle was 21 days)
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part E: TSR-042 and Carboplatin-pemetrexed
Number analyzed (Participants) | 2
Microgram per milliliter | NA (NA) — Data was not collected due to insufficient number of participants with data to calculate Cmax,ss.

186. Secondary Outcome: Part F: Cmax,ss of TSR-042
Description: as for outcome 68
Time Frame: Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed
Number analyzed (Participants) | 1
Microgram per milliliter | NA (NA) — Data was not collected due to insufficient number of participants with data to calculate Cmax,ss.

187. Secondary Outcome: Part F: Cmax,ss of TSR-022
Description: as for outcome 75
Time Frame: Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed
Number analyzed (Participants) | 1
Microgram per milliliter | NA (NA) — Data was not collected due to insufficient number of participants with data to calculate Cmax,ss.

188. Secondary Outcome: Part G: Cmax,ss of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part G.
Arm/Group | Main Study: Part G: TSR-042 and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

189. Secondary Outcome: Part H: Cmax,ss of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part H.
Arm/Group | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

190. Secondary Outcome: Part H: Cmax,ss of TSR-022
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part H.
Arm/Group | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

191. Secondary Outcome: Part I: Cmax,ss of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part I.
Arm/Group | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel
Number analyzed (Participants) | 0

192. Secondary Outcome: Part I: Cmax,ss of TSR-022
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part I.
Arm/Group | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel
Number analyzed (Participants) | 0

193. Secondary Outcome: Part A: Time to Reach Maximum Plasma Concentration (Tmax) of Niraparib
Description: as for outcome 70
Time Frame: Cycle 1: Pre-dose, 1, 2, 4, 6, 8 and 24 hours post-dose (each cycle was 21 days)
Population: PK Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD
Number analyzed (Participants) | 15 | 6
Hours | 2.250 [1.75 to 7.02] | 4.083 [2.02 to 25.65]

194. Secondary Outcome: Part A: Tmax of TSR-042
Description: as for outcome 68
Time Frame: Cycle 1: Pre-dose, 0.5, 2, 24, 96, 168, 336 and 504 hours post-dose (each cycle was 21 days)
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD
Number analyzed (Participants) | 16 | 6
Hours | 0.817 [0.50 to 2.58] | 1.750 [0.50 to 23.17]

195. Secondary Outcome: Part B: Tmax of TSR-042
Description: as for outcome 68
Time Frame: Cycle 1: Pre-dose, 0.5, 2, 24, 96, 168, 336 and 504 hours post-dose (each cycle was 21 days)
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Main Study: Part B: TSR-042 and Carboplatin-paclitaxel
Number analyzed (Participants) | 14
Hours | 1.000 [0.55 to 27.28]

196. Secondary Outcome: Part C: Tmax of Niraparib
Description: as for outcome 70
Time Frame: Cycle 1: Pre-dose, 1, 2, 4, 6, 8 and 24 hours post-dose (each cycle was 21 days)
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab
Number analyzed (Participants) | 6 | 7
Hours | 3.975 [2.00 to 23.33] | 4.050 [2.05 to 22.60]

197. Secondary Outcome: Part C: Tmax of TSR-042
Description: as for outcome 68
Time Frame: Cycle 1: Pre-dose, 0.5, 2, 24, 96, 168, 336 and 504 hours post-dose (each cycle was 21 days)
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab
Number analyzed (Participants) | 6 | 7
Hours | 1.200 [0.50 to 4.48] | 0.583 [0.50 to 2.35]

198. Secondary Outcome: Part D: Tmax of TSR-042
Description: as for outcome 68
Time Frame: Cycle 1: Pre-dose, 0.5, 2, 24, 96, 168, 336 and 504 hours post-dose (each cycle was 21 days)
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Main Study: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab
Number analyzed (Participants) | 6
Hours | 1.250 [0.50 to 25.17]

199. Secondary Outcome: Part E: Tmax of TSR-042
Description: as for outcome 68
Time Frame: Cycle 1: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Main Study: Part E: TSR-042 and Carboplatin-pemetrexed
Number analyzed (Participants) | 2
Hours | NA [NA to NA] — Data was not collected due to insufficient number of participants with data to calculate Tmax.

200. Secondary Outcome: Part F: Tmax of TSR-042
Description: as for outcome 68
Time Frame: Cycle 1: Pre-dose, 0.5, 1, 2, 3, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed
Number analyzed (Participants) | 1
Hours | NA [NA to NA] — Data was not collected due to insufficient number of participants with data to calculate Tmax.

201. Secondary Outcome: Part F: Tmax of TSR-022
Description: as for outcome 75
Time Frame: Cycle 1: Pre-dose, 0.5, 1, 2, 3, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed
Number analyzed (Participants) | 1
Hours | NA [NA to NA] — Data was not collected due to insufficient number of participants with data to calculate Tmax.

202. Secondary Outcome: Part G: Tmax of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 1: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part G.
Arm/Group | Main Study: Part G: TSR-042 and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

203. Secondary Outcome: Part H: Tmax of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 1: Pre-dose, 0.5, 1, 2, 3, 24, 48, 96, 168 and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part H.
Arm/Group | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

204. Secondary Outcome: Part H: Tmax of TSR-022
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 1: Pre-dose, 0.5, 1, 2, 3, 24, 48, 96, 168 and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part H.
Arm/Group | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

205. Secondary Outcome: Part I: Tmax of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 1: Pre-dose, 0.5, 1, 2, 3, 24, 48, 96, 168 and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part I.
Arm/Group | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel
Number analyzed (Participants) | 0

206. Secondary Outcome: Part I: Tmax of TSR-022
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 1: Pre-dose, 0.5, 1, 2, 3, 24, 48, 96, 168 and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part I.
Arm/Group | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel
Number analyzed (Participants) | 0

207. Secondary Outcome: Part A: Tmax at Steady State (Tmax,ss) of Niraparib
Description: as for outcome 70
Time Frame: as for outcome 165
Population: as for outcome 67
Measure: Median (Full Range); unit: Hours
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD
Number analyzed (Participants) | 10 | 3
Hours
  Cycle 2, n=10,3 | 4.008 [1.00 to 22.68] | 2.250 [2.08 to 7.00]
  Cycle 5, n=7,0: number analyzed (Participants) | 7 | 0
  Cycle 5, n=7,0 | 2.000 [0.00 to 2.00] |
  Cycle 11, n=2,0: number analyzed (Participants) | 2 | 0
  Cycle 11, n=2,0 | 1.817 [1.75 to 1.88] |

208. Secondary Outcome: Part A: Tmax,ss of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 152
Population: as for outcome 67
Measure: Median (Full Range); unit: Hours
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD
Number analyzed (Participants) | 9 | 4
Hours
  Cycle 4, n=9,4 | 1.500 [0.50 to 2.07] | 1.300 [0.50 to 2.70]
  Cycle 5, n=8,1: number analyzed (Participants) | 8 | 1
  Cycle 5, n=8,1 | 0.625 [0.50 to 1.73] | 2.783 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual tmax,ss for this single participant.
  Cycle 11, n=5,0: number analyzed (Participants) | 5 | 0
  Cycle 11, n=5,0 | 0.567 [0.50 to 2.00] |

209. Secondary Outcome: Part B: Tmax,ss of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 152
Population: as for outcome 67
Measure: Median (Full Range); unit: Hours
Arm/Group | Main Study: Part B: TSR-042 and Carboplatin-paclitaxel
Number analyzed (Participants) | 10
Hours
  Cycle 4, n=10 | 0.575 [0.50 to 2.08]
  Cycle 5, n=9: number analyzed (Participants) | 9
  Cycle 5, n=9 | 1.500 [0.50 to 2.10]
  Cycle 11, n=6: number analyzed (Participants) | 6
  Cycle 11, n=6 | 0.542 [0.42 to 2.07]

210. Secondary Outcome: Part C: Tmax,ss of Niraparib
Description: as for outcome 70
Time Frame: as for outcome 165
Population: as for outcome 67
Measure: Median (Full Range); unit: Hours
Arm/Group | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab
Number analyzed (Participants) | 4 | 4
Hours
  Cycle 2, n=4,4 | 4.950 [2.03 to 22.30] | 3.958 [2.00 to 6.00]
  Cycle 5, n=4,3: number analyzed (Participants) | 4 | 3
  Cycle 5, n=4,3 | 2.158 [1.82 to 2.68] | 1.967 [1.17 to 2.00]
  Cycle 11, n=3,1: number analyzed (Participants) | 3 | 1
  Cycle 11, n=3,1 | 2.000 [0.00 to 2.00] | 2.083 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual tmax,ss for this single participant.

211. Secondary Outcome: Part C: Tmax,ss of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 152
Population: as for outcome 67
Measure: Median (Full Range); unit: Hours
Arm/Group | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab
Number analyzed (Participants) | 5 | 7
Hours
  Cycle 4, n=5,7 | 1.517 [0.50 to 20.67] | 0.617 [0.50 to 2.00]
  Cycle 5, n=5,6: number analyzed (Participants) | 5 | 6
  Cycle 5, n=5,6 | 2.083 [0.50 to 2.58] | 0.825 [0.50 to 2.25]
  Cycle 11, n=4,2: number analyzed (Participants) | 4 | 2
  Cycle 11, n=4,2 | 2.000 [1.98 to 2.00] | 2.417 [2.17 to 2.67]

212. Secondary Outcome: Part D: Tmax,ss of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 152
Population: as for outcome 67
Measure: Median (Full Range); unit: Hours
Arm/Group | Main Study: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab
Number analyzed (Participants) | 5
Hours
  Cycle 4, n=5 | 0.500 [0.50 to 2.00]
  Cycle 5, n=5 | 0.550 [0.50 to 2.00]
  Cycle 11, n=4: number analyzed (Participants) | 4
  Cycle 11, n=4 | 0.500 [0.50 to 0.50]

213. Secondary Outcome: Part E: Tmax,ss of TSR-042
Description: as for outcome 68
Time Frame: Cycle 2: Pre-dose (each cycle was 21 days)
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Main Study: Part E: TSR-042 and Carboplatin-pemetrexed
Number analyzed (Participants) | 2
Hours | NA [NA to NA] — Data was not collected due to insufficient number of participants with data to calculate Tmax,ss.

214. Secondary Outcome: Part F: Tmax,ss of TSR-042
Description: as for outcome 68
Time Frame: Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed
Number analyzed (Participants) | 1
Hours | NA [NA to NA] — Data was not collected due to insufficient number of participants with data to calculate Tmax,ss.

215. Secondary Outcome: Part F: Tmax,ss of TSR-022
Description: as for outcome 75
Time Frame: Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed
Number analyzed (Participants) | 1
Hours | NA [NA to NA] — Data was not collected due to insufficient number of participants with data to calculate Tmax,ss.

216. Secondary Outcome: Part G: Tmax,ss of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part G.
Arm/Group | Main Study: Part G: TSR-042 and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

217. Secondary Outcome: Part H: Tmax,ss of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part H.
Arm/Group | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

218. Secondary Outcome: Part H: Tmax,ss of TSR-022
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part H.
Arm/Group | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

219. Secondary Outcome: Part I: Tmax,ss of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part I.
Arm/Group | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel
Number analyzed (Participants) | 0

220. Secondary Outcome: Part I: Tmax,ss of TSR-022
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part I.
Arm/Group | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel
Number analyzed (Participants) | 0

221. Secondary Outcome: Part A: Volume of Distribution After Intravenous Administration (Vss) of of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 152
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD
Number analyzed (Participants) | 8 | 2
Liter
  Cycle 4, n=5,2: number analyzed (Participants) | 5 | 2
  Cycle 4, n=5,2 | 5.5647 (1.36694) | 9.8680 (NA) — Standard deviation was not calculated as it is not statistically meaningful as there are only 2 participants.
  Cycle 5, n=8,1: number analyzed (Participants) | 8 | 1
  Cycle 5, n=8,1 | 6.6580 (1.53521) | 5.9659 (NA) — Standard deviation could not be calculated for single participant.
  Cycle 11, n=4,0: number analyzed (Participants) | 4 | 0
  Cycle 11, n=4,0 | 7.3107 (0.96007) |

222. Secondary Outcome: Part B: Vss of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 152
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Main Study: Part B: TSR-042 and Carboplatin-paclitaxel
Number analyzed (Participants) | 10
Liter
  Cycle 4, n=10 | 5.1893 (1.80311)
  Cycle 5, n=8: number analyzed (Participants) | 8
  Cycle 5, n=8 | 6.7701 (2.31992)
  Cycle 11, n=6: number analyzed (Participants) | 6
  Cycle 11, n=6 | 7.4351 (2.78481)

223. Secondary Outcome: Part C: Vss of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 152
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab
Number analyzed (Participants) | 5 | 6
Liter
  Cycle 4, n=5,5: number analyzed (Participants) | 5 | 5
  Cycle 4, n=5,5 | 6.4567 (2.68944) | 5.5177 (2.39652)
  Cycle 5, n=4,6: number analyzed (Participants) | 4 | 6
  Cycle 5, n=4,6 | 6.2405 (1.79539) | 4.8035 (0.72905)
  Cycle 11, n=4,2: number analyzed (Participants) | 4 | 2
  Cycle 11, n=4,2 | 8.9478 (3.05769) | 7.7750 (NA) — Standard deviation was not calculated as it is not statistically meaningful as there are only 2 participants.

224. Secondary Outcome: Part D: Vss of TSR-042
Description: as for outcome 68
Time Frame: as for outcome 152
Population: as for outcome 67
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Main Study: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab
Number analyzed (Participants) | 5
Liter
  Cycle 4, n=5 | 5.1493 (1.58340)
  Cycle 5, n=5 | 5.6399 (1.41478)
  Cycle 11, n=3: number analyzed (Participants) | 3
  Cycle 11, n=3 | 8.0614 (0.48037)

225. Secondary Outcome: Part E: Vss of TSR-042
Description: as for outcome 68
Time Frame: Cycle 2: Pre-dose (each cycle was 21 days)
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Main Study: Part E: TSR-042 and Carboplatin-pemetrexed
Number analyzed (Participants) | 2
Liter | NA (NA) — Data was not collected due to insufficient number of participants with data to calculate Vss.

226. Secondary Outcome: Part F: Vss of TSR-042
Description: as for outcome 68
Time Frame: Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed
Number analyzed (Participants) | 1
Liter | NA (NA) — Data was not collected due to insufficient number of participants with data to calculate Vss.

227. Secondary Outcome: Part F: Vss of TSR-022
Description: as for outcome 75
Time Frame: Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed
Number analyzed (Participants) | 1
Liter | NA (NA) — Data was not collected due to insufficient number of participants with data to calculate Vss.

228. Secondary Outcome: Part G: Vss of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part G.
Arm/Group | Main Study: Part G: TSR-042 and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

229. Secondary Outcome: Part H: Vss of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part H.
Arm/Group | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

230. Secondary Outcome: Part H: Vss of TSR-022
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part H.
Arm/Group | Main Study: Part H: TSR-042, TSR-022, and Carboplatin-nab-paclitaxel
Number analyzed (Participants) | 0

231. Secondary Outcome: Part I: Vss of TSR-042
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part I.
Arm/Group | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel
Number analyzed (Participants) | 0

232. Secondary Outcome: Part I: Vss of TSR-022
Description: Blood samples were planned to be collected at indicated time points.
Time Frame: Cycle 2: Pre-dose; Cycle 5: Pre-dose, 0.5, 2, 24, 48, 96, 168, and 336 hours post-dose (each cycle was 21 days)
Population: PK Population. Data was not collected as no participants were enrolled in Part I.
Arm/Group | Main Study: Part I: TSR-042, TSR-022, and Carboplatin-paclitaxel
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious TEAEs and STEAEs were collected up to 28.5 months in Parts A; up to 66 months in Part B; up to 60 months in Part C; up to 62.5 months in Part D; up to 4.4 months in Part E; up to 3.5 months in Part F of main study and up to approximately 19 months for PACT phase.
Description: Safety Population consisted of all participants who received any amount of study treatment. Data is presented for Parts A to F only as data was not collected for Parts G, H, and I. Parts G, H and I were not initiated due to business strategic reason. MedDRA version (v) used for Arm A and F was 23.0 and Arm B to E is 25.0.
Arm/Group | Main Study: Part A: TSR-042 and Niraparib 200 mg QD | Main Study: Part A: TSR-042 and Niraparib 300 mg QD | Main Study: Part B: TSR-042 and Carboplatin-paclitaxel | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab | Main Study: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab | Main Study: Part E: TSR-042 and Carboplatin-pemetrexed | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed | PACT Phase: Part B: TSR-042 and Carboplatin-paclitaxel | PACT Phase: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab
All-Cause Mortality (participants affected / at risk) | 4/16 | 4/6 | 7/14 | 2/6 | 5/7 | 1/6 | 1/2 | 0/1 | 0/2 | 1/1
Serious Adverse Events (participants affected / at risk) | 11/16 | 4/6 | 9/14 | 3/6 | 3/7 | 3/6 | 2/2 | 0/1 | 0/2 | 1/1
Other Adverse Events (participants affected / at risk) | 16/16 | 6/6 | 14/14 | 5/6 | 7/7 | 6/6 | 2/2 | 1/1 | 0/2 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Study: Part A: TSR-042 and Niraparib 200 mg QD (N=16) | Main Study: Part A: TSR-042 and Niraparib 300 mg QD (N=6) | Main Study: Part B: TSR-042 and Carboplatin-paclitaxel (N=14) | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab (N=6) | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab (N=7) | Main Study: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab (N=6) | Main Study: Part E: TSR-042 and Carboplatin-pemetrexed (N=2) | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed (N=1) | PACT Phase: Part B: TSR-042 and Carboplatin-paclitaxel (N=2) | PACT Phase: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertebral artery dissection (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General Medical Deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Study: Part A: TSR-042 and Niraparib 200 mg QD (N=16) | Main Study: Part A: TSR-042 and Niraparib 300 mg QD (N=6) | Main Study: Part B: TSR-042 and Carboplatin-paclitaxel (N=14) | Main Study: Part C: TSR-042, Niraparib 200 mg QD and Bevacizumab (N=6) | Main Study: Part C: TSR-042, Niraparib 300 mg QD and Bevacizumab (N=7) | Main Study: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab (N=6) | Main Study: Part E: TSR-042 and Carboplatin-pemetrexed (N=2) | Main Study: Part F: TSR-042, TSR-022, and Carboplatin-pemetrexed (N=1) | PACT Phase: Part B: TSR-042 and Carboplatin-paclitaxel (N=2) | PACT Phase: Part D: TSR-042, Carboplatin-paclitaxel and Bevacizumab (N=1)
Anaemia (Blood and lymphatic system disorders) | 4 (13) | 3 (9) | 10 (27) | 2 (9) | 5 (10) | 5 (10) | 2 (6) | 1 (12) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (4) | 1 (2) | 6 (9) | 1 (1) | 1 (1) | 4 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (7) | 2 (2) | 2 (3) | 2 (3) | 2 (5) | 2 (19) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dacryostenosis acquired (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ophthalmoplegia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (5) | 2 (2) | 4 (6) | 4 (4) | 4 (4) | 3 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (7) | 2 (2) | 4 (4) | 4 (21) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces hard (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertrophy of tongue papillae (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (10) | 4 (5) | 4 (4) | 3 (4) | 4 (6) | 3 (9) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (11) | 2 (2) | 2 (2) | 1 (2) | 4 (4) | 2 (4) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cyst rupture (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (4) | 3 (3) | 7 (9) | 2 (2) | 4 (4) | 4 (7) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 2 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (3) | 1 (1) | 2 (3) | 2 (2) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Temperature intolerance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial vulvovaginitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dacryocystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 4 (6) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiation injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Recall phenomenon (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 2 (5) | 2 (4) | 2 (4) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (6) | 1 (1) | 2 (5) | 0 (0) | 2 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 2 (4) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 2 (4) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood folate decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood testosterone decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breath sounds abnormal (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tri-iodothyronine decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin B12 decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 3 (6) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 2 (4) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 1 (4) | 1 (5) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 5 (6) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 3 (8) | 2 (4) | 1 (1) | 0 (0) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (8) | 0 (0) | 5 (6) | 0 (0) | 2 (2) | 3 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 4 (9) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 6 (11) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autonomic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 4 (5) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 3 (3) | 4 (5) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperreflexia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 4 (6) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device malfunction (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 2 (2) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocyturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 4 (9) | 3 (7) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus genital (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (4) | 3 (4) | 1 (1) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 1 (1) | 6 (7) | 2 (2) | 2 (3) | 3 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 8 (10) | 0 (0) | 1 (1) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (6) | 1 (2) | 3 (8) | 0 (0) | 1 (2) | 2 (4) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (3) | 1 (1) | 0 (0) | 4 (4) | 2 (2) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-08-15): https://cdn.clinicaltrials.gov/large-docs/85/NCT03307785/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/85/NCT03307785/SAP_001.pdf